

# **Clinical Trial Protocol**

| | Document Number: c17703547-05 |
|---|---|
| EudraCT No.: | 2017-002736-16 |
| BI Trial No.: | 1305-0012 |
| BI Investigational Product: | BI 1015550 |
| Title: | Safety, tolerability, and pharmacokinetics of multiple rising oral dose of BI 1015550 in patients with idiopathic pulmonary fibrosis (IPF) on no background anti-fibrotic therapy. |
| Lay title: | This study tests different doses of BI 1015550 in patients with idiopathic pulmonary fibrosis (IPF). The study tests how BI 1015550 is taken up by the body and how well it is tolerated. |
| Clinical Phase: | Ic |
| Clinical Trial Leader: | |
| | Phone: |
| Co-ordinating<br>Investigator: | |
| | Phone: |
| Status: | Final Protocol (Revised protocol (based on Global Amendment 4)) |
| Version and Date: | Version: 5.0 Date: 27 Mar 2019 |
| | Proprietary confidential information m International GmbH or one or more of its affiliated companies. All rights reserved l or in part - be passed on, reproduced, published or otherwise used without prior written permission |

c17703547-05  Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **CLINICAL TRIAL PROTOCOL SYNOPSIS**

| Name of company: | | Tabulated<br>Trial Protocol | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished produ | ict: | | |
| Not applicable | | | |
| Name of active ingredic | ent: | | |
| BI 1015550 | | | |
| Protocol date: | Trial number: | | Revision date: |
| 02 Nov 2017 | 1305-0012 | | 27 Mar 2019 |
| Title of trial: | | pharmacokinetics of multiple rising ic pulmonary fibrosis (IPF) on no ba | |
| Co-ordinating<br>Investigator: | | | |
| | Phone: | - <u></u> | |
| Trial site(s): | Multi-Centre study | | |
| Clinical phase: | Ic | | |
| Objectives: | Multiple Rising Dose (MRD) | | |
| | The primary objective is to investigate safety and tolerability of BI 1015550 in patients with IPF. | | |
| | The secondary objective | es are to investigate the effect of BI<br>he pharmacokinetic | 1015550 on<br>s (PK) of BI 1015550. |
| Methodology: | Double-blind, randomise design | ed within dose groups, placebo-cont | rolled, parallel-group |
| No. of patients: | | | |
| total entered: | N= 24 | | |
| each treatment: | DG 1A*: 9 (6 on active 2 on placebo) | drug and 3 on placebo) plus addition | nal 6 (4 on active drug and |
| | DG 1B*: 9 (6 on active | drug and 3 on placebo) | |
| | dose range on the basis of o | be entered to allow for testing of addition<br>experience gained during the trial conductor<br>of patients entered may exceed 18 | |
| Diagnosis: | Idiopathic Pulmonary Fi | ibrosis | |
| Main criteria<br>for inclusion: | Patients with IPF ages ≥40 years, who have not been treated with nintedanib or pirfenidone within 30 days of visit 1 and not planning to be initiated on nintedanib or pirfenidone for the duration of the study. | | |
| Test product: | BI 1015550 as tablet formulation (TF 1 containing 6mg of BI 1015550) | | |
| dose: | Starting dose of 18mg b | .i.d | |

c17703547-05 Trial Protocol


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Name of company: | | Tabulated<br>Trial Protocol | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished produ | ct: | | |
| Not applicable | | | |
| Name of active ingredie | nt: | | |
| BI 1015550 | | | |
| Protocol date: | Trial number: | | Revision date: |
| 02 Nov 2017 | 1305-0012 | 1305-0012 27 Mar 2019 | |
| mode of admin.: | Oral | Oral | |
| Reference Product | e Product Matching placebo as tablet formulation | | |
| dose: | Not applicable | | |
| mode of admin.: | mode of admin.: Oral | | |
| <b>Duration of treatment:</b> | 4 weeks | | |
| Criteria for | Secondary endpoint: | | |
| pharmacokinetics: | BI 1015550 | | |
| | Day 1: $AUC_{\tau,1}$ and $C$ | | |
| | Day 14: $AUC_{\tau,ss}$ and | $C_{max,ss}$ | |
| Criteria for safety: | Primary endpoint | | |
| | | erability of BI 1015550 by the numb | er (%) of patients with |
| | drug-related adverse eve | ents (AEs) on-treatment. | |
| | Further criteria of interest: Treatment emergent AEs (TEAEs) (including clinically elevant findings from the physical examination), safety laboratory tests (including esting for fecal occult blood and fecal calprotectin, urinalysis for hematuria), 12-lead electrocardiogram (ECG), vital signs (blood pressure (BP), pulse rate (PR), espiratory rate (RR), oral body temperature and body weight), and suicidality nonitoring. | | |
| Statistical methods: | Descriptive statistics wil | ll be calculated for all endpoints. | |

c17703547-05 Trial Protocol


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **FLOW CHART**

# Flow chart 1A: Overview

| Trial Period | Screening | | Treatment | | | | | | | End of<br>Trial | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 1 | 2 | 3 | } <sup>1</sup> | 4 | 5 | 6 | 7 | 81 | 9/<br>EOT<br>17 | T | End of<br>Trial |
| Day | -28 to -2 | -1 | 1 | 2 | 4<br>± 1 | 7<br>± 1 | 10<br>± 1 | 13 | 14 | 28<br>± 4 | | +7<br>+3 |
| Visit type | 0 | 0 | | I | 0 | 0 | 0 | 0 | V | 0 | C <sup>2</sup> | 0 |
| Informed consent | X | | | | | | | | | | | |
| Demographics <sup>3</sup> | X | | | | | | | | | | | |
| Body Weight | X | X | | | | | | | X | X | | |
| Medical History | X | X | | | | | | | | | | |
| Physical Examination | X | X | | | | | | | X | X | | X |
| Vital Signs <sup>4</sup> | X | X | X | X | X | X | X | X | X | X | | X |
| Safety Laboratory test <sup>5</sup> | X | $X^6$ | | X | X | X | X | X | | X | | X |
| Fecal Occult blood/ | X | X | | X | | X | | | X | X | | X |
| Fecal Calprotectin | | | | | | | | | | | | |
| Drug Screen/ Alcohol breath test | | X | | | | | | | | | | |
| ECG | X | X | X | X | X | X | X | | X | X | | X |

| Suicide Questionnaire <sup>8</sup> | X | X | | | | | | | X | X | X |
|---|---|---|---|---|---|---|---|---|---|---|---|
| HRCT <sup>9</sup> | X | | | | | | | | | | |
| Review of | X | X | | | | | | | | | |
| in/exclusion criteria | | | | | | | | | | | |
| Randomisation | | | X | | | | | | | | |
| BI 1015550 dispensed | | | X | X | X | X | X | X | X | | |
| BI 1015550 | | | X | X | X | X | X | X | $X^{10}$ | | |
| administration in | | | 10 | 10 | 11 | 11 | 11 | 11 | | | |
| clinic | | | | | | | | | | | |
| BI 1015550 returned | | | | | X | X | X | X | | X | |
| Compliance Check | | | | | X | X | X | X | | X | |
| Dispense diary | | | X | | X | X | X | X | | | |
| Review diary | | | | | X | X | X | X | | X | |
| PK Plasma: BI<br>1015550 | | | X<br>12 | X<br>13 | X<br>13 | | X<br>13 | X<br>13 | X 12 | X 13 | |

| Concomitant therapy | X | X | X | X | X | X | X | X | X | X | X | X | I |
|---------------------|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | 1 |


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **Footnotes Flow chart 1A**

- 1. Please refer to <u>flow chart 1B</u> and <u>flow chart 1C</u> for specifics pertaining to these visits.
- 2. Daily phone calls between study visits to assess and collect AE and confirm compliance until Day 14, with weekly phone calls between study visits thereafter until end of treatment (EOT).
- 3. Demographics (including determination of height, smoking status and alcohol history)
- 4. Vital signs include BP, PR, RR, body temperature.
- 5. Safety laboratory tests to be taken pre morning dose.
- 6. Safety laboratory tests to be taken and to be medically evaluated within 3 days prior to first administration of study drug at visit 3; this safety laboratory can be omitted, if the screening examination is performed on Days -3 or -2
- 7. DLCO is required at screening to confirm eligibility. For scheduling reasons, DLCO may be performed during or shortly following visit 1, providing results are available for review at visit 2.
- 8. Prospective suicidality monitoring, will be performed throughout this trial using the Columbia Suicidal Severity Rating scale (C-SSRS). Refer to section 5.2.5.3 and appendix 10.1 for additional details.
- 9. IPF diagnosis may be confirmed using a historical HRCT scan. If a historical scan taken within the past 12 months is not available, or an available scan fails to meet the required image acquisition specification, an HRCT may be performed after consent to determine eligibility. All HRCT scans will be sent to a central vendor for review and confirmation of IPF diagnosis, prior to randomization. HRCT should not be repeated for eligibility if previous scan was taken within the past 3 months.
- 10. All applicable doses to be administered in clinic
- 11. Morning dose to be administered in clinic
- 12. On day 1 and day 14, PK sample for BI 1015550 to be taken pre morning dose and at 0.5, 1, 1.5, 2, 4, 6, 8, 12h post dose; 12 h sample should be immediately prior to the evening dose.
- 13. PK sample for BI 1015550 to be taken pre morning dose in the morning on Days 2, 4, 10, and day 13. At day 28, PK sample to be taken ~12h post day 27 evening dose.

17. EOT visit is required for all patients, including patients who discontinue treatment early.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Flow chart 1B: Visit 3

c17703547-05

| Visit | Day | Planned time (relative to first drug<br>administration<br> h:min | Approximate clock time of actual day [h:min] | Event and comment | Safety laboratory | BI 1015550 PK blood | |
|---|---|---|---|---|---|---|---|
| | | -2:00 | 6:00-<br>8:00 | Randomization | | x <sup>1</sup> | |
| | | -0:30 | 07:30 | Breakfast | | | - |
| | | 0:00 | 08:00 | First study drug administration | | | - |
| | | 0:30 | 08:30 | | | X | - |
| | | 1:00 | 09:00 | | | $\mathbf{x}^2$ | |
| | | 1:30 | 09:30 | | | X | |
| | 1 | 2:00 | 10:00 | 240 mL fluid intake <sup>2</sup> | | X | |
| | | 4:00 | 12:00 | 240 mL fluid intake, thereafter lunch <sup>2</sup> | | Х | |
| | | 6:00 | 14:00 | | | $\mathbf{x}^2$ | - |
| 3 | | 8:00 | 16:00 | Snack (voluntary) <sup>2</sup> | | Х | |
| | | 10:00 | 18:00 | Dinner | | | |
| | | 12:00 | 20:00 | Study drug administration | | x <sup>2</sup> , | |
| | | 23:30 | 7:30 | Breakfast <sup>2</sup> | X | X | _ |
| | | 24:00 | 08:00 | Study drug administration | | | |
| | 2 | 28:00 | 12:00 | 240 mL fluid intake, thereafter lunch <sup>2</sup> | | | |
| | | 34:00 | 18:00 | Dinner | | | Ī - |
| | | 36:00 | 20:00 | Study drug administration | | | |
| | | 38:00 | 22:00 | Discharge from trial site | | | |

| Fecal occult blood and fecal calprotectin testing | | x 12-lead ECG | Vital signs | A Questioning for AEs and concomitant therapy | × Other trial procedures <sup>6</sup> |
|---|---|---|---|---|---|
| | _ | x <sup>1, 5</sup> | x <sup>1</sup> | x <sup>1</sup> | X |
| | <u> </u> | | | X | |
| | | | | А | |
| | <u> </u> | 5 | | | |
| | _ | x <sup>5</sup> | X | X | |
| | _ | x <sup>5</sup> | Х | X | |
| | | x <sup>5</sup> | Х | Х | |
| | _ | <b>x</b> <sup>5</sup> | Х | X | |
| | _ | x <sup>5</sup> | X<br>X | X<br>X | |
| | | x <sup>3,5</sup> | x <sup>3</sup> | Х | |
| X | <u> </u> | x <sup>5</sup> | X | X | |
| | | Х | X | Х | |
| | | X | X | X | |

c17703547-05

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Flow chart 1C: Visit 8

| Visit | Day | Planned time (relative to<br>first drug administration<br>[h:min] | Approximate clock time of actual day [h:min] | Event and comment | BI 1015550 PK blood | Fecal occult blood and fecal calprotectin testing |
|---|---|---|---|---|---|---|
| 8 | 14 | 311:30 | 07:30 | Breakfast <sup>2</sup> | x <sup>3</sup> | X <sup>4</sup> |
| | | 312:00 | 08:00 | Study drug administration | | |
| | | 312:30 | 08:30 | | X | |
| | | 313:00 | 09:00 | | $\mathbf{x}^2$ | |
| | | 313:30 | 09:30 | | X | |
| | | 314:00 | 10:00 | 240 mL fluid intake <sup>2</sup> | X | |
| | | 316:00 | 12:00 | 240 mL fluid intake,<br>thereafter lunch <sup>2</sup> | X | |
| | | 318:00 | 14:00 | | X | |
| | | 320:00 | 16:00 | Snack (voluntary) <sup>2</sup> | X | |
| | | 322:00 | 18:00 | Dinner | | |
| | | 324:00 | 20:00 | Study Drug administration | x <sup>2,3</sup> | |

| X 12-lead ECG <sup>5</sup> | × Vital signs | X X Questioning for AEs and concomitant therapy | × Other trial procedures 6 |
|---|---|---|---|
| X | X | X | X |
| | | X | |
| X | X | X | |
| X | X | X | |
| X | X | X | |
| X<br>X | X | X | |
| X | X | X | |
| x <sup>3</sup> | x <sup>3</sup> | X | |

#### Footnotes (flow chart 1B and 1C)

- 1. The time is approximate; the respective procedure is to be performed and completed within 2 h prior to drug administration. Allocation to treatment may be performed at any time following enrolment but must be completed prior to (first) drug administration.
- 2. If several actions are indicated at the same time point, venipuncture should be the last of the measurements and the intake of meals will be the last action.
- 3. Samples will be taken just before administration of dose.
- 4. Fecal occult blood and fecal calprotectin testing for visit 8 may be taken within 3 days of day 14 (i.e day 12-14).
- 5. The ECG recording has to be performed as triple at these time points. At baseline (i.e. Day 1, prior to drug administration) 3 triplicate ECGs are recorded within approximately one hour. The recordings should be separated by at least 15 minutes.
- 6. Other trial procedures to be performed during the visit as outlined in <u>flow chart 1A</u>.

c17703547-05 Tri

# **Trial Protocol**


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# TABLE OF CONTENTS

| TIT | LE | PAGE | 1 |
|---|---|---|---|
| CLI | INIC | AL TRIAL PROTOCOL SYNOPSIS | 2 |
| FL. | )W | CHART | 4 |
| | | OF CONTENTS | |
| | | VIATIONS | |
| 1. | INT | RODUCTION | |
| | 1.1 | MEDICAL BACKGROUND | |
| | 1.2 | DRUG PROFILE | 15 |
| | | 1.2.3 Toxicology | 16 |
| | | 1.2.5 Clinical experience in humans | 18 |
| | | 1.2.5.1 Clinical Safety | |
| | | 1.2.5.1.1 Single-Rising Dose (SRD) Study (1305.1) | |
| | | 1.2.5.1.2 Multiple-Rising Dose (MRD) study (1305.2) | 19 |
| | | 1.2.5.1.3 SRD and MRD study (1305-0011) (completed) [c22991937-01] | |
| | | 1.2.5.1.4 Food Effect (1305-0020) (completed) | |
| | | 1.2.5.1.5 Clinical experience with other PDE4 inhibitors | |
| | | 1.2.5.2 Clinical pharmacokinetics | 22 |
| | | 1.2.5.2.2 Multiple-rising dose trial (1305.2 and 1305.11, part 2) | |
| | | 1.2.5.2.3 Food effect trial (1305.20) [c20307414-01] | |
| | | 1.2.5.2.4 Prediction of human therapeutic dose range | |
| | | 1.2.6 Drug product | 25 |
| 2. | | ΓΙΟΝΑLE, OBJECTIVES, AND BENEFIT - RISK | |
| | ASS | SESSMENT | |
| | 2.1 | RATIONALE FOR PERFORMING THE TRIAL | |
| | 2.2 | | |
| | 2.3 | BENEFIT - RISK ASSESSMENT | 26 |
| | | 2.3.1 Procedure-related risks | 27 |
| | | 2.3.2 Drug-related risks and safety measures | 28 |
| | | 2.3.3 Safety measures | <b>2</b> 9 |
| <b>3.</b> | DES | SCRIPTION OF DESIGN AND TRIAL POPULATION | 31 |
| | 3.1 | OVERALL TRIAL DESIGN AND PLAN | 31 |
| | | 3.1.1 Administrative structure of the trial | 34 |
| | 3.2 | DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF | |
| | | CONTROL GROUP | 35 |

**5.2** 

| Page | 9 | of | 1 | 11 |
|------|---|----|---|----|

| 1//0354/-05 | I riai Protocoi | Page 9 of 1 |
|---|---|---|
| Proprietary confidential infor | mation © 2019 Boehringer Ingelheim International | GmbH or one or more of its affiliated companies |

| | TRF<br>4.1 | 3.3.1<br>3.3.2<br>3.3.3<br>3.3.4<br>3.3.5 | Main diagnosis for study entry Inclusion criteria Exclusion criteria Removal of patients from therapy or assessments 3.3.4.1 Removal of individual patients 3.3.4.2 Stopping criteria for dose escalation 3.3.4.3 Discontinuation of the trial by the sponsor Replacement of patients | 36<br>38<br>38<br>39 |
|---|---|---|---|---|
| | | 3.3.3<br>3.3.4<br>3.3.5 | Exclusion criteria Removal of patients from therapy or assessments 3.3.4.1 Removal of individual patients 3.3.4.2 Stopping criteria for dose escalation. 3.3.4.3 Discontinuation of the trial by the sponsor. | 37<br>38<br>39<br>40 |
| | | 3.3.4 | Removal of patients from therapy or assessments | 38<br>38<br>39 |
| | | 3.3.5 | <ul> <li>3.3.4.1 Removal of individual patients</li> <li>3.3.4.2 Stopping criteria for dose escalation</li> <li>3.3.4.3 Discontinuation of the trial by the sponsor</li> </ul> | 38<br>39<br>40 |
| | | | 3.3.4.2 Stopping criteria for dose escalation | 39<br>40 |
| | | | 3.3.4.3 Discontinuation of the trial by the sponsor | 40 |
| | | | 3.3.4.3 Discontinuation of the trial by the sponsor | 40 |
| | | | Replacement of patients | 40 |
| | | CATMI | | 4U |
| 2 | 4.1 | 11 N H TANK | ENTS | |
| | | TREA | TMENTS TO BE ADMINISTERED | 41 |
| | | 4.1.1 | Identity of BI investigational product and comparator product. | 41 |
| | | 4.1.2 | Method of assigning patients to treatment groups | 41 |
| | | 4.1.3 | Selection of doses in the trial | |
| | | | 4.1.3.1 Maximum acceptable systemic exposure, and exposure | |
| | | | multiples of selected doses | 42 |
| | | 4.1.4 | Drug assignment, dispensing and administration of doses for | |
| | | | each patient | |
| | | | 4.1.4.1 Drug Assignment | |
| | | | 4.1.4.2 Dispensing of medication | 44 |
| | | | 4.1.4.3 Administration of Doses | |
| | | 4.1.5 | Blinding and procedures for unblinding | |
| | | | 4.1.5.1 Blinding | |
| | | | 4.1.5.2 Procedures for (emergency) unblinding | |
| | | 4.1.6 | Packaging, labelling, and re-supply | |
| | | 4.1.7 | Storage conditions | 47 |
| | | 4.1.8 | Drug accountability | 47 |
| 4 | 4.2 | | COMITANT THERAPY, RESTRICTIONS, AND RESCUE | 40 |
| | | | TMENT | |
| | | 4.2.1 | Rescue medication, emergency procedures, and additional | |
| | | | treatments | |
| | | 4.2.2 | 4.2.1.1 Management of acute IPF exacerbations | |
| | | 4.2.2 | | |
| | | | 4.2.2.1 Restrictions regarding concomitant treatment | |
| | 4.0 | | 4.2.2.2 Restrictions on diet and life style | |
| | 4.3 | | TMENT COMPLIANCE | |
| <b>5.</b> ' | VAI | RIABL | ES AND THEIR ASSESSMENT | 51 |

SAFETY.......52

**6.** 

**7.** 

c17703547-05 Trial Protocol

| Page | 10 | Λf | 11 | 1 |
|-------|----|----|-----|---|
| I agu | 10 | UΙ | T 1 | L |

| Proprietary confidential | information © 2019 Boe | hrınger İngelheim İnterna | tional GmbH or one or m | ore of its affiliated companies |
|---|---|---|---|---|

| | 5.2.1 | 1 | |
|---|---|---|---|
| | 5.2.2 | | |
| | | 5.2.2.1 Definitions of adverse events | |
| | | 5.2.2.2 Adverse event collection and reporting | |
| | 5.2.3 | Assessment of safety laboratory parameters | |
| | 5.2.4 | Electrocardiogram | |
| | | 5.2.4.1 12-lead resting ECG | |
| | 5.2.5 | Assessment of other safety parameters | |
| | | 5.2.5.1 Vital signs | |
| | | 5.2.5.2 Medical examinations | |
| | | 5.2.5.3 Suicidal risk assessed by the C-SSRS | 63 |
| 5.4 | APPR | OPRIATENESS OF MEASUREMENTS | 63 |
| 5.5 | | G CONCENTRATION MEASUREMENTS AND | |
| 3.3 | | RMACOKINETICS | 64 |
| | 5.5.1 | | |
| | 3.3.1 | 5.5.1.1 Secondary endpoints | |
| | | 5.5.1.1 Secondary endpoints | |
| | 5.5.2 | Methods of sample collection | 65 |
| | 0,0,1 | 5.5.2.1 Plasma sampling for pharmacokinetic analysis | |
| | 5.5.3 | Analytical determinations | |
| | | 5.5.3.1 Analytical determination of plasma concentrations | |
| INV | /ESTIC | GATIONAL PLAN | 70 |
| 6.1 | VISIT | SCHEDULE | 70 |
| 6.2 | | ILS OF TRIAL PROCEDURES AT SELECTED VISITS | |
| 0.2 | 6.2.1 | Screening and run-in period(s) | |
| | 6.2.2 | Treatment period | |
| | 6.2.3 | Follow-up period and end of trial | |
| CT. | | CAL METHODS AND DETERMINATION OF | 1 4 |
| | | | =- |
| | | SIZE | |
| <b>7.1</b> | | ISTICAL DESIGN - MODEL | |
| | 7.1.1 | Objectives | 73 |

7.5

| - | 4 4 | • | 4 | 4 | - |
|-------|-----|----|---|---|---|
| Page | | Λt | • | | |
| 1 agc | 11 | UI | _ | 1 | _ |

| <b>7.2</b> | NULL AND ALTERNATIVE HYPOT | THESES73 |
|------------|---------------------------------------|---------------|
| <b>7.3</b> | PLANNED ANALYSES | 73 |
| | 7.3.1 Primary analyses | 73 |
| | 7.3.2 Secondary analyses | 74 |
| | 7.3.3 Safety analyses | 75 |
| | 7.3.4 Interim analyses | 76 |
| | 7.3.5 Pharmacokinetic analyses | 77 |
| 7.4 | HANDLING OF MISSING DATA | 78 |
| | 7.4.1 Safety | 78 |
| | 7.4.2 Plasma drug concentration - tip | me profiles78 |

| | <b>7.6</b> | DETERMINATION OF SAMPLE SIZE | 78 |
|---|---|---|---|
| 8. | INF | ORMED CONSENT, DATA PROTECTION, TRIAL | |
| | REC | CORDS | 80 |
| | 8.1 | STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT | |
| | <b>8.2</b> | DATA QUALITY ASSURANCE | 8 |
| | 8.3 | RECORDS | <b>8</b> 1 |
| | | 8.3.1 Source documents | <b>8</b> 1 |
| | | 8.3.2 Direct access to source data and documents | <b>8</b> 1 |
| | 8.4 | LISTEDNESS AND EXPEDITED REPORTING OF ADVERSE EVENTS | <b>8</b> 1 |
| | | 8.4.1 Listedness | 8 |
| | | 8.4.2 Expedited reporting to health authorities and IECs/IRBs | 8 |
| | 8.5 | STATEMENT OF CONFIDENTIALITY | <b>8</b> 1 |
| | <b>8.6</b> | COMPLETION OF TRIAL | 82 |
| 9. | REF | TERENCES | 83 |
| | 9.1 | PUBLISHED REFERENCES | 83 |
| | 9.2 | UNPUBLISHED REFERENCES | |
| 10. | APP | ENDICES | 87 |
| | 10.1 | COLUMBIA SUICIDAL SEVERITY RATING SCALE (C-SSRS) | 8 |

**Boehringer Ingelheim** BI Trial No.: 1305-0012

c17703547-05

27 Mar 2019

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**Trial Protocol** 

#### **ABBREVIATIONS**

ΑE Adverse event

**AESI** Adverse events of special interest

**ANCOVA** Analysis of Covariance

Area under the concentration-time curve of the analyte in plasma over a  $AUC_{\tau,1}$ 

uniform dosing interval  $\tau$  after administration of the first dose

 $AUC_{\tau,ss}$ Area under the concentration-time curve of the analyte in plasma at steady

state over a uniform dosing interval τ

ΒI Boehringer Ingelheim

b.i.d. twice daily

Below limit of quantification BLQ

BP Blood pressure

CA Competent authority CK Creatine Kinase

C-SSRS Columbia-suicide severity rating scale

CTR Clinical trial report

Maximum measured concentration of the analyte in plasma at steady state  $C_{\text{max.ss}}$ 

over a uniform dosing interval τ

Maximum measured concentration of the analyte in plasma  $C_{max}$ 

CML Local clinical monitor Central nervous system CNS

Chronic obstructive pulmonary disease **COPD** 


Boehringer Ingelheim 27 Mar 2019

BI Trial No.: 1305-0012

c17703547-05 Trial Protocol 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

CRA Clinical research associate

CRF Case report form
CRP C-reactive protein
CTP Clinical trial protocol
CTR Clinical trial report

DILI Drug induced liver impairment

ECG Electrocardiogram
EDC Electronic data capture

EDTA Ethylenediaminetetraacetic acid

EOT End of treatment FC Fecal Calprotectin

GI Gastro-intestinal gMean Geometric mean

HPLC-MS/MS High performance liquid chromatography with tandem mass spectrometry

HRCT High-resolution computed tomography

HR Heart rate

ICH-GCP ICH Harmonised Tripartite Guideline for Good Clinical Practice

IEC Independent Ethics Committee
 IPF Idiopathic Pulmonary Fibrosis
 IRB Institutional Review Board
 IRT Interactive Response Technology

ISF Investigator Site file

MedDRA Medical Dictionary for Drug Regulatory Activities

MetID A blank sample for metabolic analysis

MRD Multiple-rising dose

NC Not calculated

NIMP Non-investigational medicinal product

nM Nanomolar NOA Not analysed

NOAEL No observed adverse effect level

NOR No valid result
NOS No sample available
PD Pharmacodynamic(s)
PDE4 B Phosphodiesterase 4 B

PK Pharmacokinetic(s)

PKS Pharmacokinetic set/ parameter analysis set

PR Pulse rate

PV Pharmacovigilance

q.d. once daily

Boehringer Ingelheim 27 Mar 2019

BI Trial No.: 1305-0012

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

QT Time between start of the Q-wave and the end of the T-wave in an

electrocardiogram

QT or QT interval corrected for heart rate using the method of Fridericia (QTcF)

or Bazett (QTcB)

REP Residual effect period RR Respiratory Rate SAE Serious adverse event

SOP Standard operating procedure

SRD Single-rising dose

SUSAR Suspected Unexpected Serious Adverse Reaction

TEAEs Treatment emergent adverse events

t.i.d. three times daily

TMF Trial master file

TDMAP Trial Data Management and Analysis Plan

TSAP Trial statistical analysis plan ULN Upper limit of normal

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1. INTRODUCTION

BI 1015550 is a selective inhibitor of the Phosphodiesterase 4 B (PDE4 B) with broad anti-inflammatory and anti-fibrotic activities. It is under development for the treatment of idiopathic pulmonary fibrosis (IPF).

#### 1.1 MEDICAL BACKGROUND

Idiopathic Pulmonary Fibrosis is a specific form of chronic, progressive fibrosing interstitial pneumonia of unknown cause, occurring primarily in older adults, limited to the lungs, and associated with the histopathologic and/or radiologic pattern of usual interstitial pneumonia [P11-07084]. IPF is the most common of the 7 idiopathic interstitial pneumonias. It is a rare and fatal disease, with a median survival time of 2 to 3 years following diagnosis [R12-5527], [P11-07084]. The natural history of IPF is variable and unpredictable [R11-2587]. Disease progression is manifested by increasing respiratory symptoms, worsening pulmonary function test results, acute respiratory decline, and death.

Nintedanib and pirfenidone are the only drugs registered for the treatment of IPF and recommended in the recent ATS/ERS/JRS/ALAT Clinical Practice Guideline for the Treatment of Idiopathic Pulmonary Fibrosis [P15-07539]. Despite the availability of these drugs, the medical need remains high in this devastating disease.

BI 1015550 is a selective inhibitor of the PDE4 B with broad anti-inflammatory and anti-fibrotic activities. Based on its mode of action, BI 1015550 is hypothesized to have complementary activity to current therapies in IPF, as well as improved tolerability compared to other marketed PDE-4 inhibitors due to lower affinity for PDE4 D.

For further information, please refer to the Investigator's Brochure [c02094779-03].

#### 1.2 DRUG PROFILE

For details on nonclinical pharmacology, refer to section 5.1 in the IB [c02094779-03].


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1.2.3 Toxicology

The toxicology data support administration of BI 1015550 to women of non-child bearing potential and to men for up to 13 weeks.

The toxicity profile for BI 1015550 has been assessed in safety pharmacology studies, genetic toxicology studies, and repeat dose toxicity studies in the rat and minipig of up to 13 weeks including:

- Repeat dose toxicity studies in the rat
  - o 4 weeks (dose groups 0.2-6/12 mg/kg/day), and 13 weeks (dose groups 3-9 mg/kg/day) with 4 weeks recovery
- Repeat dose toxicity studies in the minipig
  - o 2 weeks (3-30 mg/kg/day, 2 week recovery) and 13 weeks (3-20 mg/kg/day, 4 week recovery)

Overall, vasculopathy and mortality secondary to vasculopathy are the primary findings defining the no observed adverse effect level (NOAEL) in the rat and minipig and are consistent with findings from other known PDE4 inhibitors [R10-1559]. Vasculopathy in toxicology species is thought to be a consequence of vascular tone dysregulation and subsequent inflammatory response [R17-0158]. Areas affected by vasculopathy are dependent on the nonclinical species tested. The GI tract/mesentery has been shown to be affected in multiple species (rats, minipigs, monkey) after administration of PDE4 inhibitors, including marketed compounds apremilast and roflumilast [R17-0915], [R17-0916], [R17-0919]. Additional target organs/tissues of PDE4 inhibitors include heart, liver, lung, thymus, and pancreas, and PDE4 inhibitors effects have been noted in male and female reproductive tracts of nonclinical species such as the mouse, rat, hamster, dog and monkey. Vasculopathy is considered reversible, as demonstrated in a longitudinal study performed in mice with apremilast, which showed the recovery of PDE4 inhibitor-related vasculopathy following repeated administration over 90 days [R17-0919].

Moreover, despite the observed effects in nonclinical species, two PDE4 inhibitors are used clinically and vascular injury has not been documented in humans.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

PDEi-related effects on the testes and uterus have been reported for previously marketed PDE inhibitors [R17-0915], [R17-0919].

Both marketed PDE4 inhibitors have demonstrated adverse effects in preclinical reproductive toxicity studies that include embryotoxicity or fetotoxicity and are labelled accordingly [R17-0915], [R17-0919]. Specific studies to evaluate the potential for BI 1015550 to affect male and female fertility and developmental toxicity have not yet been conducted. Therefore, adequate contraception as detailed in <u>Section 3.3.3</u> is required.

For further information please refer to the IB [c02094779-03]


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1.2.5 Clinical experience in humans

#### 1.2.5.1 Clinical Safety

Four clinical trials have been completed with BI 1015550 in healthy male volunteers:

- a single rising dose First-in-Men trial (1305.1) [U13-1792-01]
- a multiple rising dose trial (1305.2) [c02191718-02]
- a single rising dose/multiple rising dose trial (1305.11)
- a food effect trial (1305.20) [c20307414-01]

### 1.2.5.1.1 Single-Rising Dose (SRD) Study (1305.1)

BI 1015550 (0.02 mg, 0.06 mg, 0.2 mg, 0.6 mg, 2 mg, 4 mg, 8 mg, 16 mg and 24 mg dose levels) has been tested in 70 healthy male subjects. Sixteen subjects received placebo and 54 received BI 1015550. There were no notable differences between the dose groups with respect to safety and tolerability.

A total of 41 treatment emergent adverse events (TEAEs) were reported by 27 (39%) subjects. Five of these subjects (31%) received placebo. Nine subjects (12.9%) reported TEAEs that were considered drug-related by the investigator. These include drug-related diarrhea (N=3), abdominal pain (N=3), headache (N=2), and nausea/vomiting/fatigue/oral herpes in 1 subject. There was no correlation of the administered drug-dose and the number of subjects reporting at least 1 TEAE. Four of the subjects (including one subjects on placebo) reported moderate TEAEs. All subjects were reported to have recovered from TEAEs by the end-of-study examination.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

There were no suspected unexpected serious adverse reaction (SUSAR), nor any significant (based upon ICH E3), severe, serious or fatal AEs. No subject was discontinued due to AEs. In addition, no clinically relevant laboratory, vital signs and ECG changes were observed following administration of single doses of BI 1015550.

Further details can be found in IB [c02094779-03].

# 1.2.5.1.2 Multiple-Rising Dose (MRD) study (1305.2)

BI 1015550 (1 mg and 6 mg b.i.d. for two weeks) has been tested in 24 healthy male subjects. Six subjects received placebo and 18 received BI 1015550.

A total of 10 TEAEs were reported by 6 (25%) patients, 1 patient in the placebo group, 4 patients in the 1 mg group and 1 patient in the 6 mg group. The most frequent TEAEs, all of mild intensity, occurred within the CNS and GI organ classes. Reported TEAEs included headache, mild diarrhea, abdominal pain, aphtous stomatitis, mild constipation and abdominal pain. There were no GI TEAE reported in the placebo group.

Two patients were discontinued, one for personal reasons in the 1 mg b.i.d. group and one due to TEAEs in the 6 mg b.i.d. group. The latter discontinuation occurred on study Day 12 because of adverse events that were considered drug-related by the investigator. All TEAEs in this patient were of mild intensity, with the exception of C-reactive protein (CRP) increase which was of moderate intensity. Apart from the CRP increase of moderate intensity, described above, no clinically relevant laboratory findings or clinically relevant changes in vital signs or ECGs were observed following administration of repeated doses of BI 1015550.

There were no TEAEs of severe intensity, SUSARS, severe, serious or fatal AEs.

# 1.2.5.1.3 SRD and MRD study (1305-0011) (completed) [c22991937-01]

This partially randomized within dose groups, placebo-controlled trial investigated the safety, tolerability, and pharmacokinetics of single and multiple rising oral doses of BI 1015550 as tablet formulation and is an extension of the previous trials 1305.1 and 1305.2. The investigation of single (36 mg and 48 mg) and multiple (6 mg b.i.d. and 12 mg b.i.d) rising doses of BI 1015550 beyond the doses tested in the previous two trials is supported by new toxicological investigations of BI 1015550. In Part 1, BI 1015550 (36 mg and 48 mg single dose levels) was tested in 18 healthy male subjects in a partially randomised, placebo-controlled within dose groups design. Following completion of the SRD part, BI 1015550 (6 mg and 12 mg b.i.d. for two weeks) was tested in 24 healthy male subjects in a randomised, double-blind, placebo-controlled within dose groups study.

Boehringer Ingelheim BI Trial No.: 1305-0012

c17703547-05 Trial Protocol

27 Mar 2019


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c17703547-05 Trial Protocol


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For further details, see 'Investigator's Brochure' [c02094779-03].

# 1.2.5.1.4 Food Effect (1305-0020) (completed)

This open-label, randomized two-sequence, two-period crossover trial investigated the relative bioavailability of BI 1015550 following oral administration of 24 mg BI 1015550 under fed and fasted conditions. Twelve (12) healthy male subjects were entered.

[c20307414-01].

#### 1.2.5.1.5 Clinical experience with other PDE4 inhibitors

Selective PDE4 inhibitors have been approved for chronic obstructive pulmonary disease (COPD) with chronic bronchitis and a history of exacerbations (roflumilast), and for moderate to severe plaque psoriasis and active psoriatic arthritis (apremilast). Roflumilast has been tested in Phase III studies for asthma and apremilast in Phase III studies for active Behcet's disease. No PDE4 inhibitor has been tested in IPF, yet.

#### **Cilomilast**

Cilomilast was the first selective PDE4 inhibitor developed for the maintenance of lung function (forced expiratory volume in one second (FEV1)) in patients with COPD but failed to demonstrate efficacy to support approval of the drug. Cilomilast nonclinical findings


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

include mesenteric arteritis in rats. In the clinical program the frequency of GI AEs was high. Fecal occult blood testing was benign with unremarkable colonoscopy findings in the few patients with blood in the stool. Lack of approval was based on inadequate evidence of efficacy rather than any safety concern [P06-08316].

#### Roflumilast

This PDE4 inhibitor (Daxas® in EU, Daliresp® in US) got approved for treatment of COPD. More than 5,000 patients with COPD were included in the "COPD Safety Pool". The most frequently reported AEs associated with roflumilast treatment were GI events (diarrhea, weight loss, nausea, abdominal pain) and headache followed by insomnia, dizziness and decreased appetite. There was an increased incidence of neuropsychiatric adverse reactions such as insomnia, anxiety, nervousness and depression; in rare instances suicidal ideation behavior (including completed suicide). Atrial fibrillation as SAE was reported more often in patients treated with

roflumilast. Among the AEs leading to death, cardiac arrest was reported in a higher number of patients who received roflumilast [R10-1555]. Clinical manifestation of mesenteric vasculitis, an adverse effect that has been a concern with PDE4 inhibition in general, was not reported in these clinical studies.

#### Apremilast

One PDE4 inhibitor for treatment of active psoriatic arthritis (Otezla®) has been approved by the FDA for moderate to severe plaque psoriasis. Otezla® has been evaluated in 1493 patients with active psoriatic arthritis in three randomized placebo-controlled studies [R17-1427] Access date 29, March 2017.). The most common adverse reactions were diarrhea, headache and nausea, followed by vomiting, upper respiratory tract infection, nasopharyngitis and abdominal pain. The product information of Otezla® recommends the close monitoring of patient's body weight and its cautious use in patients with history of depression and/or suicidal thoughts or behavior [R14-1795].

Boehringer Ingelheim BI Trial No.: 1305-0012 c17703547-05

27 Mar 2019

Trial Protocol


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1.2.5.2.2 Multiple-rising dose trial (1305.2 and 1305.11, part 2)

Pharmacokinetics of BI 1015550 was investigated in healthy male volunteers given multiple oral doses of 1 mg and 6 mg b.i.d. with solution formulation in a fasted condition (Study 1305.2) and 6 and 12 mg bid with tablet formulation in a fed condition (Study 1305.11).

27 Mar 2019

**Trial Protocol** 


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1.2.5.2.3 Food effect trial (1305.20) [c20307414-01]

A two-way crossover, single dose, food effect study (24 mg, N=12) was performed.

# 1.2.5.2.4 Prediction of human therapeutic dose range

Observed target engagement data in the previous clinical trials [<u>U13-1792-01</u>] and [<u>c02191718-02</u>] supported by population pharmacokinetic-pharmacodynamic (PK-PD) modelling predicts a human therapeutic dose range of 12 mg - 24 mg BI 1015550 b.i.d. The


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

estimated exposure at these doses range from free maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval  $\tau$  (free  $C_{max,ss}$  of 81.1 nM and free AUC<sub>0-24,ss</sub> of 1072 nM·h at the 12 mg bid dose to free  $C_{max,ss}$  of 193 nM and free AUC<sub>0-24,ss</sub> of 1983 nM·h at 24 mg b.i.d., respectively). These exposures are below the target maximum exposure margin for humans of 277 nM (free  $C_{max,ss}$ ) and 2284 nM·h (free AUC<sub>0-24,ss</sub>) based on the 13-week rat study (section 4.1.3.1).

# 1.2.6 Drug product

BI 1015550 is a non-hygroscopic, white to off-white to light yellow powder. It is a poorly soluble compound with high permeability.

For further details, see 'Investigator's Brochure' [c02094779-03].

c17703547-05


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 2. RATIONALE, OBJECTIVES, AND BENEFIT - RISK ASSESSMENT

#### 2.1 RATIONALE FOR PERFORMING THE TRIAL

Based on the limitations of the current therapy of IPF there is a medical need to slow or halt the progression of this disease (see <u>section 1.1</u>). BI 1015550 is a selective PDE4 B inhibitor with a pleiotropic and broad mode of action (MoA) that has the potential to offer improved efficacy and/or tolerability as add-on to registered anti-fibrotics or as a mono therapy in IPF.

As the planned doses to be tested fall within the estimated therapeutic range and based on the safety profile of this class of compound, the safety, tolerability and PK of rising doses of BI 1015550 will be evaluated in IPF patients.

The current design will provide essential information for clinical development of BI 1015550 as a treatment for IPF with the aim of determining the optimal dose of BI 1015550 based on PK, safety and tolerability.

#### 2.2 TRIAL OBJECTIVES

with IPF.

Description of the endpoints to be determined, and the observations along with specific information as how to collect the data for that information, is provided in <u>section 5</u>.

The primary objective is to investigate safety and tolerability of BI 1015550 in patients with IPF. The secondary objectives are to

evaluate the pharmacokinetics (PK) of BI 1015550 in patients

#### 2.3 BENEFIT - RISK ASSESSMENT

Experiments have shown that BI 1015550 affects the fibrotic pathway and the effects may be complementary and synergistic to those of nintedanib. It is postulated that BI 1015550 may provide therapeutic benefit to patients with lung fibrosis, but this has not yet been shown clinically [c02094779-03]. Patient participation in the study is of major importance to investigate the safety, tolerability and PK profile of BI 1015550.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Based on study 1305.11 using indirect target engagement in healthy volunteers at single doses up to 48 mg q.d., therapeutic efficacy might be expected from 12 mg b.i.d but may not plateau at that dose. Given the morbidity associated with IPF, dose escalation within the therapeutic range in a patient population rather than healthy subjects is considered acceptable to also assess target engagement in the relevant population. Given the morbidity associated with IPF, dose escalation within the therapeutic range in a patient population rather than healthy subjects is considered acceptable. The expected exposure at the planned doses of 18 mg b.i.d and 24 mg b.i.d fall within range of the estimated therapeutic range and are below the pre-defined maximal acceptable human systemic exposure limit. As such, the benefit-risk of these doses in a patient population is considered positive. Accordingly, dose escalation within the current protocol starting with administration of 18 mg b.i.d will be assessed in IPF patients. Evaluation of the 12 mg b.i.d dose, which has been evaluated in healthy volunteers (1305.11), will only be performed in this study if the safety and tolerability of the 18 mg b.i.d dose is not supported.

Furthermore, given the potential overlap in tolerability profile between BI 1015550 and the currently approved standard of care for IPF, dose escalation will be performed on no background therapy in order to adequately evaluate the tolerability and safety profile of the compound. To mitigate potential risk associated with a placebo controlled study in this patient population, only patients not currently treated with anti-fibrotic or not planned to be treated within 4 weeks of Visit 3 will be targeted for participation. Initiation of treatment for management of acute deterioration will be allowed at any time during the study at the discretion of the treating physician.

The patients are exposed to the risks of the study procedures and the risks related to the exposure to the trial medication (see section 2.3.1).

It is hypothesized that BI 1015550 will ultimately lead to improved efficacy and an acceptable tolerability profile, resulting in a positive benefit/risk profile.

#### 2.3.1 Procedure-related risks

The use of an indwelling venous catheter for the purpose of blood sampling may be accompanied by mild bruising and also, in rare cases, by transient inflammation of the wall of the vein. In addition, in rare cases a nerve might be injured while inserting the venous catheter, potentially resulting in paresthesia, reduced sensibility, and/or pain for an indefinite period. The same risks apply to venipuncture for blood sampling.

ECG electrodes may cause local and typically transient skin reactions.

The total volume of blood withdrawn during the entire study will not exceed 400 mL per patient over the duration of the trial. This is less than the volume of a normal blood donation (500 mL). No health-related risk to the patients is expected from this blood withdrawal.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 2.3.2 Drug-related risks and safety measures

There are no listed adverse events or expected events defined for BI 1015550 based on the available data.

BI 1015550 is considered a low risk compound for the purpose of this trial based on the following observations:

- BI 1015550 has been used in humans before (although in lower doses) and was considered safe and well-tolerated
- BI 1015550 is not a first in class compound. Other PDE4-inhibitors have been previously evaluated by other companies and two are approved (see <u>section 1.2.5.1.5</u>)
- Both rat and minipig are considered relevant species for BI 1015550 with toxicology data showing the rat as the most sensitive species [c02094779-03].
- The nature of the target and the mechanism of action of BI 1015550 are well understood [c02094779-03].

Below is a summary of the known safety profile for the PDE4 class of compounds:

Vasculopathy: Vasculopathy is a typical side effect of PDE4 inhibitors in rats.

The predicted exposure for the doses to be tested in the current study falls below the maximum tolerable limit set based on the NOAEL.

As there are no validated biomarkers for vasculitis, routine monitoring of surrogate markers as performed in previous PDE-4 programs will be done as part of standard safety assessment including:

- Hematology panel (to detect changes by bleeding or inflammation)
- Inflammation markers (hsCRP, fibrinogen, erythrocyte sedimentation rate (ESR), fecal calprotectin)
- Immunochemical based fecal occult blood test as a sensitive method to detect occult blood in the stool
- Urinalysis (dipstick to detect hematuria followed by urine microscopy in case of positive results)

Of note, safety monitoring as described above was suggestive of an inflammatory process in the GI tract of one subject in trial 1305.2, where moderate elevation in CRP was observed. At the same time, the subject developed mild GI-AEs (section 1.2.5.1.2). The subject was therefore discontinued from study drug administration.

Safety monitoring continued showing normalization within days and the subject recovered.

*Emesis and further GI adverse events:* 

Based on the two completed clinical trials [<u>U13-1792-01</u>] and [<u>c02191718-02</u>] BI 1015550 was generally well tolerated at the doses tested with only mild to moderate GI side effects.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

<u>Depression and Suicidality</u>: Apremilast and roflumilast, two of the currently marketed PDE4 inhibitors, are associated with increased risk of depression with some patients reporting suicidal ideation and attempts and also reported cases of completed suicide. Accordingly, symptoms of depression and suicidality will be monitored using the Columbia-suicide severity ranking score (C-SSRS). If a patient exhibits serious suicidality in the clinical judgment of the investigator or according to the C-SSRS, assessment the patient will be discontinued (for details refer to <u>section 3.3.4.1</u> and <u>appendix 10.1</u>).

<u>Reproductive toxicity</u>: PDEi-related effects on the testes have been shown nonclinically for the marketed compounds ampremilast and roflumilast (section 1.2.5.1.5).

Developmental and reproductive studies have not yet been conducted; therefore the effect of sub therapeutic concentrations of BI 1015550 or its metabolites with regards to embryofetal risk has not been explored. In order to address this risk, patients will be informed accordingly and be required to use adequate contraception as detailed in <u>section 3.3.3.</u>

# 2.3.3 Safety measures

Although rare, a potential for drug-induced liver injury is under constant surveillance by sponsors and regulators. Therefore, this study requires timely detection, evaluation, and follow-up of alterations in selected liver laboratory parameters to ensure patients' safety. See also <u>section 5.2.2.1</u>, adverse events of special interest.

The following precautionary measures will be taken in this study in order to minimize the risk for patients:

- Careful dose selection as described in <u>section 4.1.3</u>. For each group, patients will be divided into two cohorts. The first cohort will consist of 3 patients (2 on active and 1 on placebo), the second of 6 patients (4 on active, 2 on placebo). Within each dose level, the two cohorts will be separated by at least 72 hours (between 1st patients of each cohort)
- A maximum acceptable human exposure has been defined based on toxicity findings (see section 4.1.3.1).
- Dose escalation will be guided by measurements of BI 1015550 (free C<sub>max</sub> and free AUC<sub>0-24,ss</sub>). Prior to each dose escalation, the estimated systemic exposure of the next higher dose group will be calculated using PK data from the preceding dose group to ensure that the estimated exposure does not exceed the pre-defined maximum acceptable human exposure limit.
- Decision for dose escalation will be made after blinded review of the data by the safety review committee (see <u>section 3.1.1</u> and <u>section 4.1.5.2</u>), in a documented Safety Review meeting which will take place after all patients in the first dose group


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

(18mg b.i.d, group 1A) have completed 14 days of treatment. Dose escalation to 24 mg b.i.d. is only permitted if both safety/tolerabilty (from all 9 patients) and PK projections (from a minimum of 4 patients on active treatment) are acceptable and if none of the pre-specified stopping criteria are met (section 3.3.4). The minimum time interval between last patient completing dosing at day 14 in the first cohort of a given dose group and the first dosing in the next higher dose group is 7 days. For details see section 3.1 and section 3.3.4.

- Safety laboratory examinations including surrogate markers of inflammation/vasculitis will be performed as described in section 2.3.2.
- Repeated single and triple 12-lead ECGs during inpatient PK visits will be performed.
- During inpatient visits, the patients will be under medical observation and thoroughly monitored for both expected and unexpected adverse events.
- Male Subjects have to use adequate contraception as detailed in <u>section 3.3.3</u> and female subjects of childbearing potential are not eligible to participate.

After completing the first 14 days of treatment, the appropriateness of the patients to remain and continue treatment will be done by PI or delegate based on continued assessment of benefit-risk profile for each patient.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3. DESCRIPTION OF DESIGN AND TRIAL POPULATION

#### 3.1 OVERALL TRIAL DESIGN AND PLAN

This study will test multiple doses of BI 1015550. For a schematic overview, refer to <u>figure</u> 3.1:1.

Figure 3.1:1 1305-0012 Study Design Overview



This trial is double-blind, randomised, and placebo-controlled within parallel dose groups. A total of 18 male and female patients with IPF are planned to participate in 2 sequential groups consisting of 9 patients per group. However, additional patients may be entered to allow testing of additional doses within the planned dose range on the basis of results obtained from the 1305-0011 trial as well as experience gained during trial conduct (e.g. preliminary PK data), provided the planned and approved highest dose will not be exceeded. Thus, the actual number of patients entered may exceed 18, but will not exceed 30 patients entered. Such changes may be implemented via non-substantial clinical trial protocol (CTP) amendments\*\*.

Within each dose group, 6 patients will receive the active drug and 3 will receive placebo. Only one dose is tested within each dose group. Each dose group will consist of 2 cohorts which will be treated subsequently for safety reasons as outlined in section 2.3.3.

\*\*An additional 6 patients (4 on active, 2 on placebo) will be entered in dose group 1A (18mg bid)

The first 36 hours of drug administration will be done in an inpatient setting to monitor for any acute reaction. Patients will then be treated outpatient with daily follow up by study

c17703547-05

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

personnel by telephone, and interim clinic visits for monitoring during the first 14 days. Thereafter, patients will be contacted weekly by telephone, for monitoring with interim clinic visits until 4 weeks. This monitoring schedule was selected in order to optimize feasibility and based on known safety profile of this class of compound which are primarily limited to GI tolerability in clinical studies.

For a schematic overview of design and decision points, refer to <u>figure 3.1:2</u>.

Figure 3.1:2 Design and decision point



The dose groups to be evaluated are outlined in <u>Table 3.1: 1</u>. Patients will take medication twice daily, for the duration of the trial.

Table 3.1: 1 Dose groups

| Dose Group | 1. | A | 1B* | |
|---|---|---|---|---|
| Dose Level | 0 | | -1 | 1 |
| Daily Dose (mg) | 36 | | 24 | 48 |
| Dose Regimen | 18 mg b.i.d | | 12 mg b.i.d | 24 mg b.i.d |
| Number of patients | 9 6** | | 9 | 9 |
| Patients receiving placebo | 3 | 4 | 3 | 3 |
| Patients receiving active drug | 6 | 2 | 6 | 6 |

\*The daily dose for group IB may be reduced to 24 mg delivered as 12 mg b.i.d dosing regimen, if the safety, tolerability or PK profile of the 18 mg b.i.d dose is determined to be unacceptable.

<sup>\*\*</sup> An additional 6 patients (4 on active, 2 on placebo) will be entered in dose group 1A (18mg bid). A documented safety review meeting will take place to review the full 18mg bid group data (9 + 6 patients), prior to dose escalation.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The dose groups (group 1A and group 1B) will be investigated consecutively, maintaining a time interval of at least 7 days between the last patient completing dosing at day 14 in the previous dose group and the first drug administration of the subsequent dose group.

A documented safety review meeting will take place prior to dose escalation. The decision to escalate the dose will be made by the sponsor after consultation with the safety review committee (see section 3.1.1) based on in-depth analysis of all available safety data, especially SAEs (if occurred), AEs and out-of-range laboratory results (if considered clinically significant) and PK data (from a minimum of 4 patients on active treatment). Safety Reviews may be conducted face-to-face or by video/telephone conference. The clinical trial leader is responsible for organization and minutes of the reviews. A summary will be filed in the ISF at each site and in trial master file (TMF).

- The dose will be escalated to 24 mg b.i.d if no safety concerns arose in the preceding dose group (i.e. no dose-limiting events occurred) and if none of the pre-specified trial-specific stopping criteria were met (refer to section 3.3.4.2).
- In the event the 18 mg b.i.d dose is found to have acceptable safety but an unacceptable PK projection for 24 mg, the second dose group 1B will be cancelled.
- In the event the 18 mg b.i.d dose is determined to have unacceptable safety or tolerability, the dosing of group 1B will be reduced to 12 mg b.i.d and the patients continuing with extended treatment in the 18 mg b.i.d group 1A will be stopped. The 12 mg b.i.d dose will be used to confirm the safety and tolerability of the 12 mg b.i.d dose previously tested in healthy volunteers, in the target patient population, as well as to evaluate disease specific biomarkers over 12 weeks.

An unscheduled safety review meeting can be requested anytime for any reasonable cause by the coordinating investigator or the sponsor of the study, e.g. because of any unforeseen adverse events, etc.

The minimum data set for safety review consists of the following data:

- AEs in the current and preceding dose group (including clinically relevant findings from ancillary safety testing listed below) (Note: AEs may be ongoing at the time of Safety Reviews and AE information may be subject to change prior to Database Lock)
- Results from 12-lead EGG in the current and preceding dose groups.
- Vital signs in the current and preceding dose groups
- Clinical laboratory tests in the current and preceding dose groups
- Preliminary PK data for selected time as per section 7.3.4.
- Check of criteria for stopping patient treatment as per section 3.3.4.1

The sponsor is allowed to alter the scheduled dose levels (e.g. add an intermediate dose level) within the planned dose range on the basis of experience gained during the study. This may include PK data suggesting an exposure close to or just above predefined thresholds or initial safety signals with open causality (not dose limiting), providing the planned and approved


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

highest dose is not exceeded. In this case, the total number of patients in this trial might increase. The sponsor should stop dose escalation in case the safety evaluation leads to concerns that would not allow higher dosing.

An overview of all relevant activities is provided in the <u>Flow Charts 1A</u>, <u>1B</u>, and <u>1C</u>. For visit schedules and details of trial procedures at selected visits, refer to <u>sections 6.1</u> and <u>section</u> <u>6.2</u>, respectively.

The trial will terminate after all patients have completed the scheduled study visits or discontinue study treatment, whichever comes first.

#### 3.1.1 Administrative structure of the trial

The trial will be conducted in approximately 20 sites in Europe.

A safety review committee will be responsible for blinded review of safety and PK data in order to guide decisions pertaining to dose used in subsequent treatment groups. The safety review committee will be composed of representatives from the sponsor, the coordinating investigator as well as an external expert not otherwise involved in the trial. The committee will retain the ability to unblind patients(s) as required (refer to section 4.1.5.2). This is not expected to cause bias with regards to data assessment or analyses. Following each data safety review meeting, a meeting will be held with trial investigators to review the blinded data and discuss the recommendation from the safety review committee.

A coordinating investigator is responsible to coordinate investigators at the different sites participating in this trial. The coordinating investigator (or appropriately qualified delegate) will participate in safety review meetings and will be involved in the discussions to escalate the dose.

BI has appointed a clinical trial leader, responsible for coordinating all required activities, in order to:

- manage the trial in accordance with applicable regulations and internal standard operating procedure (SOP),
- direct the clinical trial team in the preparation, conduct, and reporting of the trial
- ensure appropriate training and information of local clinical monitors (CML), clinical research associate (CRA), and participating trial sites.

The trial medication will be provided by the Clinical Trial Supplies Unit, BI Pharma GmbH & Co. KG, Biberach, Germany.

On-site monitoring will be performed by BI or a contract research organisation appointed by BI.

Safety laboratory tests will be performed by a central laboratory appointed by BI.

The analyses of BI 1015550 in plasma will be performed at BI or a suitable contract research organization (CRO).


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The digitally recorded 12-lead ECGs will be sent to a specialized contract research organization for evaluation.

Data management and statistical evaluation will be done by BI or by a suitable contract research organization (CRO) under the responsibility of BI and according to BI SOPs.

Tasks and functions assigned in order to organize, manage, and evaluate the trial are defined according to BI SOPs. A list of responsible persons and relevant local information can be found in the ISF.

The trial is sponsored by Boehringer Ingelheim Pharma GmbH & Co. KG, Germany.

# 3.2 DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUP

For multiple-rising dose trials, the design described in <u>section 3.1</u> is viewed favourable under the provision not to expose the patients involved to undue risks since the main study objective is to investigate safety and tolerability of BI 1015550.

A double blind design is appropriate to reduce observer bias and evaluate safety and tolerability.

Given the morbidity associated with IPF, and potential differences regarding fibrotic status dose escalation within the therapeutic range in a patient population for 4 weeks rather than healthy subjects is considered acceptable. The expected exposure at the planned doses of 18 mg bid and 24 mg bid fall within range of the estimated therapeutic range and are below the pre-defined maximal acceptable human systemic exposure limit. As such, the benefit-risk of evaluating of these doses in a patient population is considered positive. Accordingly, within the current protocol dose escalation starting with administration of 18 mg b.i.d is planned in IPF patients to minimize exposure of patients to sub-therapeutic doses and build on the data already obtained in healthy volunteers at 12 mg for 2 weeks. Evaluation of the 12 mg b.i.d dose for 4 weeks is only planned in this trial if the safety and tolerability of the 18 mg b.i.d dose is not supported.

It is standard in Phase 1 trials to include a placebo group as control for the evaluation of safety and tolerability. Each dose group consists of 9 patients with 6 on active treatment, and 3 on placebo\*\*. The placebo control group includes all patients of all dose groups treated with placebo. 6 patients per active treatment group are in general considered as sufficient for the exploratory evaluation of pharmacokinetics.

\*\* An additional 6 patients (4 on active, 2 on placebo) will be entered in dose group 1A (18mg bid).

Non clinical toxicology data currently supports studies up to 12 weeks of durations. The treatment duration of 4 weeks is sufficient to capture safety and tolerability of a PDE4 inhibitor in support of longer term studies, evaluate PK and exploration of induction potential,


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Disease specific biomarkers and pulmonary function outcomes would require longer than 4 weeks. Recent disease specific biomarker data from the INMARK study (1199-0227) suggest that effects in disease specific biomarkers would require much larger sample size and with longer duration, even beyond 12 weeks to gain a robust evaluation of disease specific biomarkers. Four weeks data allows first generation of normative data on BI 1015550.

#### 3.3 SELECTION OF TRIAL POPULATION

It is planned that 18 male and female patients with a confirmed diagnosis of IPF will enter the study. The actual number of patients entered may exceed the total of 18 if additional intermediate doses will be tested (see section 3.1).

Only male patients and postmenopausal or surgically sterilised female patients will be included into the study because hitherto no data on reproductive toxicology are available.

A log of all patients enrolled into the study (i.e. having given informed consent) will be maintained in the investigator site file (ISF) at the investigational site irrespective of whether they have been treated with investigational drug or not.

Reasons for screen failures will be collected in the electronic Case Report Form (eCRF). The re-screening of screen failed patients may be permitted in certain cases after discussion with the trial team. A patient will not be permitted to re-screen more than one time and must meet inclusion/exclusion to be eligible for randomization. For patients re-screened, a new informed consent should be signed and the patient will be assigned a new unique patient number.

# 3.3.1 Main diagnosis for study entry

Patients diagnosed with IPF and who comply with eligibility requirements may qualify for participation in the trial.

#### 3.3.2 Inclusion criteria

Patients will only be included into the trial, if they meet the following criteria:

- 1. Signed and dated written informed consent prior to admission to the study in accordance with ICH Harmonised Tripartite Guideline for Good Clinical Practice (ICH-GCP) and local legislation
- 2. Male or female patients aged  $\geq$ 40 years at visit 1.
- 3. A clinical diagnosis of IPF based on ATS/ERS/JRS/ALAT 2011 guideline (P11-07084) within the previous 5 years as confirmed by the investigator based on chest high-resolution computed tomography (HRCT) scan taken within 12 months of visit 1 and confirmed by central review prior to visit 2.
- 4. Forced Vital Capacity (FVC) ≥50% of predicted normal at visit 1
- 5. Diffusion capacity of the lung for carbon monoxide (DLCO) (corrected for haemoglobin [Hb] [Visit 1]): > 30% of predicted normal at visit 1
c17703547-05

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3.3.3 Exclusion criteria

Patients will not be allowed to participate if any of the following general criteria apply:

- 1. Patients with a significant disease or condition other than IPF which in the opinion of the investigator, may put the patient at risk because of participation, interfere with study procedures, or cause concern regarding the patient's ability to participate in the study.
- 2. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
- 3. Surgery of the GI tract that could interfere with PK of the trial medication (except appendectomy).
- 4. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders including but not limited to mood disorders.
- 5. Evidence of active infection (chronic or acute) based on clinical exam or laboratory findings.
- 6. History of allergy or hypersensitivity to the trial medication or its excipients
- 7. Use of drugs within 30 days prior to administration of trial medication that are known to influence the results of the trial including time between start of the Q-wave and the end of the T-wave in an electrocardiogram (QT) / QT interval corrected for heart rate using the method of Fridericia (QTcF) or Bazett (QTcB) (QTc)
- 8. A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males or repeatedly greater than 470 ms in females) or any other relevant ECG finding at screening
- 9. A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
- 10. Participation in another trial where an investigational drug has been administered within 30 days or less than 5 half-lives (whichever is greater) of the respective drug prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug.
- 11. Inability to refrain from smoking on trial days
- 12. Alcohol abuse (consumption of more than 20 g per day)
- 13. Active drug abuse
- 14. Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
- 15. Inability to comply with dietary regimen required for the trial

Boehringer Ingelheim BI Trial No.: 1305-0012 c17703547-05

27 Mar 2019


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Trial Protocol

- 16. Patient is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
- 17. Male patients who do not agree to minimize the risk of female partners becoming pregnant from first dosing day until two months after the study completion. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive used for at least two months prior), true sexual abstinence (when this is in line with the preferred and usual lifestyle of the patient), or surgically sterilized, including vasectomy.
- 18. Females who are not surgically sterilised or who are not postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous levels of Follicle-stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory).
- 19. Relevant airways obstruction (i.e. pre-bronchodilator FEV1/FVC <0.7) at visit 1
- 20. Patients who have previously been treated with nintedanib or pirfenidone within 30 days of visit 1.
- 21. Positive fecal occult blood (no retest allowed),

22.

- 23. Positive testing for hematuria if confirmed by microscopic urine analysis (retest allowed)
- 24. Any lifetime history of suicidal behavior (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior)
- 25. Any suicidal ideation of type 2 to 5 on the C-SSRS in the past 12 months (i.e. active suicidal thought without method, intent or plan; active suicidal thought with method, but without intent or plan; active suicidal thought with method and intent but without specific plan; or active suicidal thought with method, intent and plan).

For study restrictions, refer to section 4.2.2.

#### 3.3.4 Removal of patients from therapy or assessments

#### 3.3.4.1 Removal of individual patients

An individual patient is to be removed from the trial if:

- 1. The patient withdraws consent, without the need to justify the decision
- 2. The patient needs to take concomitant drugs that interfere with the investigational product or other trial medication
- 3. The patient is no longer able to participate for other medical reasons (such as surgery, adverse events, or diseases)
- 4. An AE or clinically significant laboratory change or abnormality occurred that the investigator judges to warrant discontinuation of treatment. This may include cases of sustained symptomatic hypotension (BP <90/50 mmHg) or hypertension (BP >180/100


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

mmHg) or of clinically relevant changes in ECG requiring intervention as well as unexplained liver enzyme elevations at any time during the trial.

- 5. The patient shows an elevation of AST and/or ALT ≥3-fold upper limit of normal (ULN) combined with an elevation of total bilirubin ≥2-fold ULN (measured in the same blood sample) and/or needs to be followed up according to the drug induced liver impairment (DILI) checklist provided in the case report form (CRF).
- 6. The subject exhibits serious suicidality, in the clinical judgment of the investigator or according to the following criteria:
  - any suicidal behavior (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behaviour)
  - any suicidal ideation of type 4 or 5 in the C-SSRS (i.e. active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent)

In addition to these criteria, the physician may discontinue patients at any time based on his or her clinical judgment.

A patient can also be removed from the trial if eligibility criteria are being violated or if the patient fails to comply with the protocol (for instance, by non-adherence to dietary rules, or non-attendance at study assessments).

If a patient is removed from or withdraws from the trial after first administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF. In this case, the data will be included in the CRF/trial database and will be reported in the clinical trial report (CTR). At the time of discontinuation a complete end of trial examination will be performed if possible and the information will be recorded in the CRFs. These discontinuations will be discussed in the CTR.

## 3.3.4.2 Stopping criteria for dose escalation

Dose escalation will not proceed if

- 1. More than 50% of the patients of one dose group on active drug show drug-related and clinically relevant adverse events of moderate or severe intensity during planned safety review.
- 2. At least 2 subjects at one dose level on active drug showed relevant individual QT prolongation, i.e. a QTc increase of greater 60 ms from baseline in connection with absolute QT or QTc greater than 500 ms, which has been confirmed by a repeat ECG recording.
- 3. The measured gMean free C<sub>max</sub> or free AUC of one dose group increases above the following exposure thresholds or if the estimated gMean exposure of the next dose group is expected to exceed a free C<sub>max,ss</sub> of 277 nM or a free AUC<sub>0-24,ss</sub> of 2284 nM·h. Estimation will be done at specified time points based on preliminary PK results of preceding dose groups as specified in section 7.3.4.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3.3.4.3 Discontinuation of the trial by the sponsor

Boehringer Ingelheim reserves the right to discontinue the trial overall or at a particular trial site at any time for any of the following reasons:

- 1. New toxicological findings or serious adverse events (SAE) invalidate the earlier positive benefit-risk-assessment.
- 2. The trial will be terminated if at least one drug-related SAE is reported that is considered to be unacceptable.
- 3. The expected enrolment goals overall or at a particular trial site are not met
- 4. Violation of ICH-GCP, or the CTP, or the contract with BI by a trial site or investigator, disturbing the appropriate conduct of the trial
- 5. The sponsor decides to discontinue the further development of the investigational product.

The investigator / the trial site will be reimbursed for reasonable expenses incurred in case of trial termination (except in case of the fourth reason).

#### 3.3.5 Replacement of patients

In case some patients do not complete the trial, the clinical trial leader together with the trial pharmacokineticist and the trial statistician are to decide if and how many patients will be replaced. A replacement patient will be assigned a unique study patient number, and will be assigned to the same treatment as the patient he or she replaces.

c17703547-05 Trial Protocol 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4. TREATMENTS

#### 4.1 TREATMENTS TO BE ADMINISTERED

The investigational product has been manufactured by BI Pharma GmbH & Co. KG.

#### 4.1.1 Identity of BI investigational product and comparator product

The characteristics of the test product are given below:

Substance: BI 1015550

Pharmaceutical formulation: Tablet Formulation (TF1)

Source: BI Pharma GmbH & Co. KG, Germany

Unit strength: 6 mg

Posology: Dose group 1A: 3-0-3

Dose group 1B: 2-0-2 or 4-0-4

Route of administration: p.o.

Duration of use: 28 days b.i.d. dosing

The characteristics of the reference product (placebo) are given below:

Substance: Placebo matching in size and weight to 6 mg tablet

Pharmaceutical formulation: Tablet formulation

Source: BI Pharma GmbH & Co. KG, Germany

Unit strength: n.a.

Posology: Dose group 1A: 3-0-3

Dose group 1B: 2-0-2 or 4-0-4

Route of administration: p.o.

Duration of use: 28 days b.i.d. dosing

#### 4.1.2 Method of assigning patients to treatment groups

At the screening visit, patients will be informed about the planned visit dates. The patients willing to participate will be recruited to groups according to their temporal availability (group 1A vs group 1B).


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

At visit 3, eligible patients will be randomised to receive active drug or placebo. The randomisation will occur in a blinded fashion via Interactive Response Technology (IRT). The IRT system will assign the appropriate medication number based on the treatment allocated. The randomisation code will be controlled and documented. All instructions for use of the IRT system will be described in a user guide/ manual which will be available in the ISF.

The randomisation procedure is described in <u>section 7.5.</u>

#### 4.1.3 Selection of doses in the trial

Trial 1305-0012 is an extension of the previous multiple rising dose trial (1305-0011) and proceeds with dose escalation. The doses selected for this trial cover a lower estimated therapeutic range and fall below the maximum acceptable systemic exposure.

The recommended maximum target dose is based on an exposure multiple against the predefined maximal acceptable human systemic exposure limit. This is calculated as a ratio of the maximal acceptable human exposure (see <u>section 4.1.3.1</u>) divided by predicted systemic exposure after single dosing based on the free fraction.

A starting dose of 18 mg b.i.d. of BI 1015550 has been selected, based on safety, tolerability and PK data, as well as indirect target engagement data from the completed study 1305.11 and multiple doses

up to 12 mg bid in healthy volunteers. These data will be provided through an annually updated IB. If supported by the safety and PK data from the 18 mg b.i.d. dose group, a second dose group will be initiated at the maximum targeted dose of 24 mg b.i.d. Based on simulations incorporating pre-clinical data and data from previously conducted clinical trials, it is expected that following escalation from 18 mg b.i.d. to 24 mg b.i.d., exposure will increase in a dose proportional manner. As such, this is the highest dose where the expected systemic exposure is within the therapeutic range and below the pre-defined human maximum acceptable exposure limit (Table 4.1.3.1: 1).

A b.i.d dosing allows administration of the same daily dose with an increased safety margin with regards to Cmax. Further, a lower Cmax following b.i.d. dosing compared to q.d dosing is also assumed to lead to fewer tolerability issues.

4.1.3.1 Maximum acceptable systemic exposure, and exposure multiples of selected doses

The maximal acceptable human systemic exposure limit is derived from the primary toxicological findings of vasculopathy and mortality observed in the rat and minipig (see section 1.2.3).

Boehringer Ingelheim BI Trial No.: 1305-0012 c17703547-05 27 Mar 2019

**Trial Protocol** 


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

<u>Table 4.1.3.1:1</u> shows the predicted maximum human exposure (AUC) for the planned doses to be tested in the current protocol, all of which fall below the pre-defined human maximum acceptable exposure limit.

c17703547-05


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.1.4 Drug assignment, dispensing and administration of doses for each patient

## 4.1.4.1 Drug Assignment

The treatments to be evaluated are outlined in Table 4.1.4.1: 1 below. The number of units for placebo corresponds to the number of units of the respective dose level.

Table 4.1.4.1: 1 BI 1015550 and placebo treatments, oral administration

| Dose | Substance | Pharmaceutical form | Unit strength | Number of units per administration | Total daily dose |
|---|---|---|---|---|---|
| 1A | BI 1015550 | Tablet | 6mg | 3 tablets in the morning and evening | 36 mg |
| 1B | BI 1015550 | Tablet | 6mg | 2 or 4 tablets in the morning and evening | 24 or 48<br>mg |
| 1A-1B | Placebo* | Tablet | | Identical to active treatment | |

<sup>\*</sup> Patients receiving placebo are equally distributed across dose groups

## 4.1.4.2 Dispensing of medication

Based on the treatment allocated at randomization, the IRT system will be used to dispense the appropriate medication kits at each visit.

Medication is packaged in bottles containing 20 tablets. To ensure patients receive adequate supply of study medication, kits (bottles) will be dispensed at clinic visits in quantities as outlined in <u>table 4.1.4.2: 1</u>.

c17703547-05

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 4.1.4.2: 1 Quantity of medication kits dispensed per visit

| Visit | Day | Group 1A: 18mg b.i.d<br># bottles dispensed | Group 1B: 24mg b.i.d <sup>1</sup> # bottles dispensed | Group 1B: 12mg b.i.d <sup>1</sup> # bottles dispensed |
|---|---|---|---|---|
| 3 | 1 | 1 <sup>2</sup> | 1 <sup>2</sup> | 1 <sup>2</sup> |
| 3 | 2 | 1 | 1 | 0 |
| 4 | 4 | 2 | 2 | 1 |
| 5 | 7 | 2 | 2 | 1 |
| 6 | 10 | 2 | 2 | 1 |
| 7 | 13 | 13 | 1 <sup>3</sup> | <b>1</b> <sup>3</sup> |
| 8 | 14 | 5 | 7 | 3 |

- 1. Dose tested in group 1B will be based on safety and PK result from dose group 1A.
- 2. Patients will retain bottle dispensed at day 1, when discharged at day 2.
- 3. Patients will retain bottle dispensed at day 13, when discharged at day 14.

#### 4.1.4.3 Administration of Doses

Study Medication- BI 1015550

The first administration of trial medication will be in the clinic, at visit 3 (day 1).

When in clinic, the trial medication will be administered to the patients, while in a standing position, as an oral dose together with about 240 mL of water under supervision of the investigating physician or an authorised designee. The so-called four-eye principle (two-person rule) should be applied for administration of trial medication

During the first 2 h after drug administration, they are not allowed to lie down (i.e. no declination of the upper body of more than 45 degrees from upright posture except for medical examination), or to sleep. Patients will be kept under close medical surveillance from the morning of Day 1 to the evening of Day 2 and all day on Day 14.

To ensure a dosing interval of 12 h, the administration of trial medication should take place at the same time every morning and evening.

While at home, the trial medication should be taken at approximately the same time each morning and evening, with one glass of water.

Patients will be given a medication diary to record daily intakes of medication taken at home since the last clinic visit.

For restrictions with regard to diet see section 4.2.2.2.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 4.1.5 Blinding and procedures for unblinding

#### 4.1.5.1 Blinding

This trial is designed double-blind with regard to the patients and the investigators (as well as the research staff at the trial site) in order to eliminate observer or performance bias. This means avoiding systematic differences in assessments regarding the patient's treatment (active or placebo). According to the trial design, the current dose level will be known to patients and investigators.

At the sponsor, access to the randomisation schedule is restricted to the Clinical Trial Support group, who generates the randomisation code and labels, and to the Pharmaceutics Department, where the packaging takes place. Access to the codes will be controlled and documented by a signed confidentiality statement, which will be stored in the TMF.

Within the ECG laboratory, the staff involved with interval measurements and assessments will be blinded with respect to the treatment and also with regard to the recording date and time as well as the time points of the ECGs. The interval measurements for a given patient will be performed in a random and blinded sequence by a single technician. No more than two different blinded readers will evaluate the ECGs of the study.

If an interim safety analysis of ECG data is required, a part of the staff of the ECG laboratory may be unblinded. This part of the staff is strictly separated from those parts of the staff, which is involved with interval measurements and assessments of single ECGs (blinded).

Prior to unblinding of the trial database, the randomisation codes may be provided to bioanalytical staff/trial pharmacokineticist to perform preliminary PK analyses. The Trial Bioanalyst and trial pharmacokineticist will sign a confirmation that the codes will be treated confidentially and results will only be shared in a blinded fashion.

The trial will only be unblinded after locking of the database.

## 4.1.5.2 Procedures for (emergency) unblinding

The safety review committee (except the coordinating investigator) will retain the ability to unblind patients(s) via IRT as required to review the trial specific stopping criteria based on active treatment (see <a href="section 3.3.4.2">section 3.3.4.2</a>). By this the members of the review committee (except the coordinating investigator) will be unblinded but the unblinding information will not be distributed to other personnel involved in the study. The reason for unblinding must be documented in the minutes along with the date and initials of the person who broke the code.

Emergency unblinding will be available to the investigator/ pharmacist/ investigational drug storage manager via IRT. It must only be used in an emergency situation when the identity of the trial must be known to the investigator in order to provide appropriate medical treatment or otherwise assure safety of trial participants. The reason for unblinding must be documented in the source documents and/or appropriate CRF page, along with the date and initials of the person who broke the code.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Due to the requirements to report SUSARs, it may be necessary for a representative from BI's Pharmacovigilance (PV) group to assess the randomisation code for individual patients during trial conduct. The access to the code will only be given to authorised PV representatives and not shared further.

#### 4.1.6 Packaging, labelling, and re-supply

Drug supplies will be provided by Boehringer Ingelheim..

The investigational product will be packaged and labelled in accordance with the principles of Good Manufacturing Practice. Re-supply to the sites will be managed via an IRT system, which will also monitor expiry dates of supplies available at the sites.

For details of packaging and the description of the label, refer to the ISF.

The clinical trial supply will be packaged in bottles holding the trial medication (20 tablets per bottle), which are labelled with trial identification.

The sponsor and name, address and telephone number of the trial site are given in the patient information form. The EudraCT number is indicated on the title page of this protocol as well as on the patient information and informed consent forms. Examples of the labels will be available in the ISF.

#### 4.1.7 Storage conditions

Drug supplies will be kept in their original packaging and in a secure limited access storage area according to the recommended (labelled) storage conditions. Where necessary, a temperature log must be maintained to make certain that the drug supplies are stored at the correct temperature. If the storage conditions are found to be outside the specified range, the local clinical monitor (as provided in the list of contacts) is to be immediately contacted.

#### 4.1.8 Drug accountability

The investigator / pharmacist / investigational drug storage manager will receive the investigational drugs delivered by the sponsor when the following requirements are fulfilled:

- Approval of the study protocol by the IRB / ethics committee
- Availability of a signed and dated clinical trial contract between the sponsor and the principle investigator
- Approval/notification of the regulatory authority, e.g. competent authority
- Availability of the curriculum vitae of the principal investigator
- Availability of a signed and dated clinical trial protocol or immediately imminent signing of the clinical trial protocol.

Only authorised personnel as documented in the form 'Trial Staff List' may dispense medication to trial patients. The trial medication must be administered in the manner specified in the CTP. All unused trial medication must be returned to the sponsor. Receipt, usage and return must be documented on the respective forms. Account must be given for any discrepancies.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The investigator / pharmacist / investigational drug storage manager must maintain records of the product's delivery to the trial site, the inventory at the site, the use by each patient, and the return to the sponsor.

These records will include dates, quantities, batch / serial numbers, expiry ('use-by') dates, and the unique code numbers assigned to the investigational products and trial patients. The investigator / pharmacist / investigational drug storage manager will maintain records that document adequately that the patients were provided the doses specified by the CTP, and that reconcile all investigational products received from the sponsor. At the time of return to the sponsor (and/or) appointed CRO, the investigator / pharmacist / investigational drug storage manager must verify that all unused or partially used drug supplies have been returned by the clinical trial patient and that no remaining supplies are in the investigator's possession.

# 4.2 CONCOMITANT THERAPY, RESTRICTIONS, AND RESCUE TREATMENT

#### 4.2.1 Rescue medication, emergency procedures, and additional treatments

There are no specific rescue drugs foreseen for the treatment of AEs. No special emergency procedures are to be followed. In case of adverse events in need of treatment, the investigator can authorise symptomatic therapy. In those cases, patients will be treated as necessary and, if required, kept under supervision at the trial site or transferred to a hospital until all medical evaluation results have returned to an acceptable level.

All concomitant or rescue treatment taken during the course of the trial must be recorded in the source document and on the CRF.

#### 4.2.1.1 Management of acute IPF exacerbations

In case of acute IPF exacerbation or worsening in baseline condition, all treatment options considered adequate by the Investigator are allowed. Efforts should be made to keep the subject on study medication. Sponsor should be contacted prior to stopping study drug.

#### 4.2.2 Restrictions

#### 4.2.2.1 Restrictions regarding concomitant treatment

All concomitant or rescue therapies will be recorded (including time of intake on study days) on the appropriate pages of the CRF.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 4.2.2.1:1 Restricted medication

| Medication | Prior to<br>Study | Screening<br>Period | PK Evaluation<br>Period (Day 1-<br>14) | Extended<br>treatment<br>period<br>(Day 15+) | Follow up period |
|---|---|---|---|---|---|
| Potent p-gp<br>inhibitor or inducer | Not permitted <sup>1</sup> | Not permitted | Not permitted | Not permitted | Permitted |
| Potent and<br>moderate CYP3A<br>inhibitors or<br>inducers | Not permitted <sup>1</sup> | Not<br>permitted | Not permitted | Not permitted | Permitted |
| Nintedanib | Refer to exclusion 20 | Not permitted | Not permitted | Not permitted <sup>3</sup> | Permitted |
| Pirfenidone | Refer to exclusion 20 | Not permitted | Not permitted | Not permitted <sup>3</sup> | Permitted |
| Other anti-fibrotic therapies | Not permitted <sup>1</sup> | Not permitted | Not permitted | Not permitted | Permitted |
| PDE inhibitors <sup>2</sup> | Not permitted <sup>1</sup> | Not permitted | Not permitted | Not permitted | Permitted |
| Sensitive substrate of CYP3A | Permitted | Permitted | Use with caution | Use with caution | Permitted |

**Footnotes to restricted medication Table 4.2.2.1:1** 

- 1. Not permitted 30 days prior to randomization (visit 3)
- 2. Includes, for example: Sildenafil, tadalafil, vardenafil, roflumilast, apremilast.
- 3. Based on clinical status, standard of care treatment may be initiated prior to the end of 4 weeks, but should be avoided where possible as the safety has not been previously assessed and interference with trial related endpoints cannot be excluded. To allow for assessment of disease relevant markers at 4 weeks, use of SOC should be limited where possible.

#### 4.2.2.2 Restrictions on diet and life style

While admitted to the trial site the patients are restricted from consuming any other foods or drinks than those provided by the staff. Standardised meals will be served at the time points described in the <u>Flow Chart</u>. No food is allowed for at least 4 h after drug intake.

On PK profile days (i.e., Day 1 and Day 14) liquid intake is restricted from 1 hour before administration until lunch with exception of the fluid administered with the breakfast and the drug, and ~240 mL of water at 2 and 4 hours post-dose (mandatory for all patients). From lunch until 24 hours post-dose, water intake is restricted to 3000 mL. On PK profile days (i.e., Day 1 and Day 14), standardized meals will be served at 4, and 10 hours following drug administration. Snacks should be served at times as outlined in the flow chart.

Grapefruits, Seville oranges (sour or bitter oranges) and their juices, and dietary supplements and products including St. John's wort (Hypericum perforatum) are not permitted starting 7


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

days before the first administration of trial medication until after the last PK sample is collected.

Alcoholic beverages are not permitted starting 7 days before the first administration of trial medication until after the last PK sample is collected at day 14. After day 14 the use of alcohol should be limited but is not prohibited.

Smoking is not allowed during in-house confinement at the trial site.

Methylxanthine-containing drinks or foods (such as coffee, tea, cola, energy drinks, and chocolate) are not allowed from 24 h preceding the administration of trial medication and until the end of plasma PK sampling of the respective visit.

Excessive physical activity (such as competitive sport) should be avoided starting 7 days before the first administration of trial medication until the end of trial examination.

Direct exposure to the sun or exposure to solarium radiation should be avoided during the entire study.

#### 4.3 TREATMENT COMPLIANCE

During visits, compliance will be assured by administration of all trial medication in the study centre under supervision of the investigating physician or a designee. The measured plasma concentrations will provide additional confirmation of compliance.

Patients are requested to bring all remaining trial medication, including empty bottles with them when attending visits.

Based on tablet counts (unused), treatment compliance will be calculated as shown in the formula below. Compliance will be verified by the CRA authorised by the sponsor.

Treatment compliance % = Number of tablets actually taken x 100

Number of tablets which should have been taken

If the number of doses taken is not between 80% and 120%, site staff will explain to the patient the importance of treatment compliance.

Patients who are non-compliant (for instance, who do not appear for scheduled visits or violate trial restrictions) may be removed from the trial and the CRF will be completed accordingly (for further procedures, please see section 3.3.4.1).

c17703547-05 Trial Protocol


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5. VARIABLES AND THEIR ASSESSMENT


c17703547-05

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5.2 SAFETY

## 5.2.1 Endpoints of safety

The primary endpoint to assess safety and tolerability of BI 1015550 by the number (%) of patients with drug-related AEs on-treatment.

Further endpoints:

Further criteria of interest:

- TEAEs (including clinically relevant findings from the physical examination)
- Safety laboratory tests (including testing for fecal occult blood and fecal calprotectin and urinanalysis for hematuria)
- 12-lead ECG
- Vital signs (blood pressure, pulse rate, respiratory rate, oral body temperature and body weight)
- Suicidality monitoring

#### 5.2.2 Assessment of adverse events

#### 5.2.2.1 Definitions of adverse events

#### Adverse event

An adverse event (AE) is defined as any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a patient in a clinical investigation who received a pharmaceutical product. The event does not necessarily have to have a causal relationship with this treatment.

#### Serious adverse event

A SAE is defined as any AE which fulfils at least one of the following criteria:

- results in death,
- is immediately life-threatening, which refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if more severe,
- requires inpatient hospitalisation or
- requires prolongation of existing hospitalisation
- results in persistent or significant disability / incapacity, or
- is a congenital anomaly/birth defect, or


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

• is deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgement which may jeopardise the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions.

Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of dependency or abuse

#### AEs considered 'Always Serious'

Cancers of new histology and exacerbations of existing cancer must be classified as a serious event regardless of the duration between discontinuation of the drug and must be reported as described in <u>section 5.2.2.2</u>, subsections 'AE collection' and 'AE reporting to sponsor and timelines'.

In accordance with the European Medicines Agency initiative on Important Medical Events, Boehringer Ingelheim has set up a list of further AEs, which by their nature, can always be considered to be 'serious' even though they may not have met the criteria of an SAE as defined above.

The latest list of 'Always Serious AEs' can be found in the electronic data capture (EDC) system. These events should always be reported as SAEs as described above.

#### Suicidal Risk assessed by the C-SSRS

The C-SSRS is a semi-structured, investigator-rated interview, developed by clinical experts in cooperation with the FDA, assessing both suicidal behavior and suicidal ideation. It does not give a global score, but provides some categorical and some severity information specifically for behavior and ideation.

The C-SSRS interview may be administered by any type of physician, psychologist, clinical social worker, mental health counselor, nurse, or coordinator with C-SSRS training. It has a typical duration of five minutes, and causes only a low burden on subjects. At a minimum, the interview consists of 2 screening questions related to suicidal ideation and 4 related to suicidal behavior and may be expanded to up to 17 items in case of positive responses. Free text entries are allowed for; the investigator has to directly evaluate the scale and write a report.

The C-SSRS has been widely used in large multinational clinical trials. The C-SSRS will be administered at the screening visit (using the 'screening' version) with the aim to exclude subjects with active moderate or severe symptomatology within a specified time prior to the screening or baseline visit. The life time history of suicidal ideation and behavior will also be recorded.

After the screening/baseline visit the assessment 'since last visit' will be performed at each clinic visit ('since last visit' version).


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The investigator is to review all positive and negative reports for plausibility and clinical relevance. Doubtful reports may be validated by a consulting psychiatrist. If there is a confirmed positive report of suicidal behavior or suicidal ideation type 4 or 5 after start of trial, the investigator is to immediately interview the subject during the clinic visit and/or is to consult a psychiatrist. If the positive report is confirmed, appropriate actions for the subject's safety have to be initiated.

All C-SSRS reports of <u>suicidal ideation type 4 and 5 and all reports of suicidal behavior must</u> <u>be reported as separate SAEs by the investigator.</u>

For self-injurious behavior, no suicidal intent' standard AE/SAE reporting rules are to be applied.

For each negative report (Suicidal ideation type 1, 2 or 3) after the start of the trial, the investigator is to decide based on clinical judgement whether it represents an adverse event (AE) as defined in the protocol, and if it is considered an AE then it must be reported accordingly.

## **Adverse events of special interest (AESIs)**

The term AESI relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this trial, e.g. the potential for AEs based on knowledge from other compounds in the same class. AESIs need to be reported to the sponsor's PV Department within the same timeframe that applies to SAEs, please see above.

The following are considered as AESIs:

#### • Hepatic injury

A hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- o an elevation of AST and/or ALT ≥3 fold ULN combined with an elevation of total bilirubin ≥2 fold ULN measured in the same blood sample, and/or
- o aminotransferase (ALT, and/or AST) elevations ≥10 fold ULN

These lab findings constitute a hepatic injury alert and the patients showing these lab abnormalities need to be followed up according to the DILI checklist provided in the eCRF. In case of clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the Investigator should make sure these parameters are analysed, if necessary in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described in the DILI checklist should be followed.

#### Intensity (severity) of AEs

The intensity (severity) of the AE should be judged based on the following:

Mild: Awareness of sign(s) or symptom(s) which is/are easily tolerated Moderate: Sufficient discomfort to cause interference with usual activity

Severe: Incapacitating or causing inability to work or to perform usual activities


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### Causal relationship of AEs

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest that there is a reasonable possibility of a causal relationship could be:

- The event is consistent with the known pharmacology of the drug
- The event is known to be caused by or attributed to the drug class.
- A plausible time to onset of the event relative to the time of drug exposure.
- Evidence that the event is reproducible when the drug is re-introduced
- No medically sound alternative aetiologies that could explain the event (e.g. preexisting or concomitant diseases, or co-medications).
- The event is typically drug-related and infrequent in the general population not exposed to drugs (e.g. Stevens-Johnson syndrome).
- An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is diminished).

Arguments that may suggest that there is no reasonable possibility of a causal relationship could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident (e.g. pre-treatment cases, diagnosis of cancer or chronic disease within days / weeks of drug administration; an allergic reaction weeks after discontinuation of the drug concerned)
- Continuation of the event despite the withdrawal of the medication, taking into account the pharmacological properties of the compound (e.g. after 5 half-lives). Of note, this criterion may not be applicable to events whose time course is prolonged despite removing the original trigger.
- Additional arguments amongst those stated before, like alternative explanation (e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned).
- Disappearance of the event even though the trial drug treatment continues or remains unchanged.

#### 5.2.2.2 Adverse event collection and reporting

#### **AE Collection**

The investigator shall maintain and keep detailed records of all AES in the patient files.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The following must be collected and documented on the appropriate CRF(s) by the investigator:

- From signing the informed consent onwards until the individual patient's end of trial: -all AEs (serious and non-serious) and all AESIs.
- After the individual patient's end of trial:

The investigator does not need to actively monitor the patient for AEs but should only reported related SAEs and related AESIs of which the investigator may become aware of by any means of communication, e.g. phone call. Those AEs should however, not be reported in the CRF.



Figure 5.2.2.2:1 AE reporting requirements

The REP for BI 1015550, when measurable drug levels or PD effects are still likely to be present, is defined as 7 days after the last administration of BI 1015550. Therefore, all AEs which occurred through the treatment phase and throughout the REP will be considered as on treatment; please see Section 7.3.3. Events which occurred after the REP but prior to the last per protocol contact will be considered as follow up events.

#### AE reporting to sponsor and timelines

The investigator must report SAEs, AESIs and non-serious AEs which are relevant for the reported SAE or AESI on the BI SAE form via fax immediately (within 24 hours) to the sponsor's unique entry point (country specific contact details will be provided in the ISF). The same timelines applies if follow-up information becomes available. In specific occasions the investigator could inform the sponsor upfront via telephone. This does not replace the requirement to complete and fax the BI SAE form.

With receipt of any information to these events, a follow-up SAE form has to be provided. For follow-up information the same rules and timelines apply as for initial information.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## Information required

For each AE, the investigator should provide the information requested on the appropriate eCRF pages, and the BI SAE form, if applicable. The investigator should determine the causal relationship to the trial medication.

The following should also be recorded as an (S)AE in the CRF and BI SAE form (if applicable):

- Worsening of the underlying disease or of other pre-existing conditions
- Changes in vital signs, ECG, physical examination and laboratory test results, if they are judged clinically relevant by the investigator.

If such abnormalities already pre-exist prior to trial inclusion they will be considered as baseline conditions and should be collected in the eCRF only.

All (S)AEs, including those persisting after individual patient's end of trial must be followed up until they have resolved, have been assessed as "chronic" or "stable" or no further information can be obtained.

#### **Pregnancy**

In rare cases, pregnancy might occur in a clinical trial. Once a patient has been enrolled in the clinical trial and has taken trial medication, the investigator must report any drug exposure during pregnancy in a trial participant immediately (within 24 hours) by means of Part A of the Pregnancy Monitoring Form to the sponsor's unique entry point.

Similarly, potential drug exposure during pregnancy must be reported if a partner of a male trial participant becomes pregnant. This requires a written consent of the pregnant partner.

The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported to the sponsor's unique entry point on the Pregnancy Monitoring Form for Clinical Trials (Part B).

The ISF will contain the Pregnancy Monitoring Form for Clinical Trials (Part A and B).

As pregnancy itself is not to be reported as an AE, in the absence of an accompanying SAE and/or AESI, only the Pregnancy Monitoring Form for Clinical Trials and not the SAE Form is to be completed. If there is an SAE and/or AESI associated with the pregnancy, an SAE form must be completed in addition.

#### 5.2.3 Assessment of safety laboratory parameters

For the assessment of laboratory parameters, blood and urine samples will be collected by the trial site at the time points indicated in the <u>Flow Chart</u> after the patients have fasted for at least 10 h. Overnight fasting is not required at the discretion of the investigator or designate for retests.

The parameters that will be determined are listed in <u>Table 5.2.3: 1</u> and <u>table 5.2.3: 2</u>. Reference ranges will be provided in the ISF.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Manual differential white blood cell count or urine sediment examinations will only be performed if there is an abnormality in the automatic blood cell count or in the urinalysis, respectively, i.e. if automatic count is not feasible or differential WBC is abnormal (i.e. pathological or atypical cells) and clinically relevant in the opinion of the investigator. In case the urinalysis is positive for erythrocytes, leukocytes, nitrite or protein, microscopic examination of the urine sediment will be performed. Positive findings of the urine sediment examination will be monitored and if needed based on the medical judgment of the investigator an urologist may be consulted.

Fecal occult blood testing and fecal calprotectin testing will be performed by the central laboratory. Both tests will be performed at the time points indicated in the Flow Chart. As patients may not be able to defecate at the trial site in the morning of the visit, after screening (visit 1) they may collect the specimen at home and bring the test specimen to the trial site after the screening visit, within the screening period. In addition, samples collected within 3 days prior to first dosing (ie day -3 to day -1) may be collected as visit 2 (day -1) sample and samples collected within 3 days prior to subsequent visits may be used, with the exception of the sample taken at day 2.

In case of GI AEs (e.g. diarrhea, constipation), additional testing for fecal occult blood and fecal calprotectin may be carried out at the discretion of the investigator. If a patient tests positive for occult blood in feces, further tests will be performed and the patient will be monitored closely.

Table 5.2.3: 1 Routine laboratory tests

| Functional lab group | Test name |
|---|---|
| Haematology | Haematocrit Haemoglobin Red blood cell count (RBC) Reticulocyte count White blood cell count (WBC) Platelet count Erythrocyte sedimentation rate (ESR) |
| Automatic WBC differential (relative and absolute) | Neutrophils, eosinophils, basophils, monocytes, lymphocytes |
| Manual differential WBC (if automatic differential WBC is abnormal) Coagulation | Polymorphnuclear neutrophils (segs), band neutrophils (stabs), eosinophils, basophils, monocytes, lymphocytes Activated partial thromboplastin time (aPTT) Prothrombin time (Quick's test and INR) Fibrinogen |
| Enzymes | Aspartate transaminase (AST/GOT) Alanine transaminase (ALT/GPT) Alkaline phosphatase (AP) Gamma-glutamyl transferase (GGT) Creatine kinase (CK) CK-MB, only if CK is elevated Lactate dehydrogenase (LDH) Lipase Amylase |
| Hormones <sup>1</sup> | Thyroid stimulating hormone (TSH) fT3, fT4 |
| Substrates <sup>1</sup> | Plasma glucose Creatinine Total bilirubin Direct and indirect bilirubin Total protein High sensitivity C-Reactive Protein (hs CRP) Uric acid Total cholesterol Triglycerides |
| Electrolytes | Albumin Sodium Potassium Chloride Calcium Inorganic phosphate |

c17703547-05 Trial Protocol 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 5.2.3: 2 Exclusionary laboratory tests

| Functional lab group | Test name |
|-----------------------------|-------------------------------------------|
| Drug screening (urine) | Amphetamine/MDA |
| | Barbiturates |
| | Benzodiazepine |
| | Cannabis |
| | Cocaine |
| | Methadone |
| | Methamphetamines/MDMA/XTC |
| | Opiates |
| | Phencyclidine |
| | Tricyclic antidepressants |
| Infectious serology (blood) | Hepatitis B surface antigen (qualitative) |
| | Hepatitis B core antibody (qualitative) |
| | Hepatitis C antibodies (qualitative) |
| | HIV-1 and HIV-2 antibody (qualitative) |

The tests listed in Table 5.2.3: 2 are exclusionary laboratory tests which may be repeated as required. The results will not be entered in the CRF/database and will not be reported in the CTR. Infectious serology will be tested at screening (visit 1) only. Drug screening is to be performed at visit 2 (day -1).

To encourage compliance with alcoholic restrictions, a breath alcohol test will be performed at visit 2, and may be repeated at any time during the study at the discretion of an investigator or designate. The results will not be included in the CTR.

The laboratory tests listed in <u>Table 5.2.3: 1</u> and 5.2.3: 2 will be performed at a central lab as selected by Boehringer Ingelheim, with the exception of the drug screening, which will be performed at the trial site.

Laboratory data will be transmitted electronically from the laboratory to the trial site.

## 5.2.4 Electrocardiogram

## 5.2.4.1 12-lead resting ECG

#### Recording

Twelve-lead resting ECGs (I, II, III, aVR, aVL, aVF, V1 - V6) will be recorded using a computerised electrocardiograph which will be provided to the sites, at the time points given in the Flow Chart.

In order to achieve a stable heart rate (HR) at rest and to assure high quality recordings at comparable resting phases, all ECGs will be recorded for 10-sec duration after the patients have rested for at least 10 min in a supine position. The site personnel will be instructed to assure a relaxed and quiet environment so that all patients are at complete rest during the recordings. ECG assessment will always precede all other study procedures of the same time point (except blood drawing from an intravenous cannula which is already in place) to avoid compromising the ECG quality.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Electrode placement will be performed according to the method of Wilson, Goldberger and Einthoven or limb leads modified by Mason and Likar (hips and shoulders instead of ankles and wrists).

ECGs will be recorded as single ECGs or as triple ECGs (three single ECGs recorded within 180 sec) as indicated in the Flow Chart.

ECGs may be repeated for quality reasons for instance due to alternating current artefacts, muscle movements, or electrode dislocation. For repetition within triplicate ECGs the time window of 180 sec applies as well. The repeat ECGs are assigned to the respective scheduled time point.

Additional (unscheduled) ECGs may be recorded for safety reasons. These ECGs are assigned to the prior scheduled time point in the sponsor's database.

#### Data transfer

All ECGs will be transferred electronically to the central ECG lab for storage and evaluation.

In case of repeat ECGs due to quality reasons, all ECGs will be transferred to the central ECG lab who will select the correct one for analysis.

Unscheduled ECGs (for safety reasons) will be transferred to the central ECG lab but will not be included into the statistical analysis of interval lengths.

Data transfer from the central ECG lab to the sponsor is described in the ECG data transfer agreement (see TMF).

#### **Evaluation**

#### a) Central ECG lab

Central ECG lab evaluation will be performed for the first of three replicate ECGs per time point on Day 1, day 2 (planned time 23:30h only) and day 14. For baseline, where 3 triplicate ECGs are recorded, only the first single ECG per triplicate ECG (i.e. 3 single ECGs) will be evaluated.

This will include the determination of cardiac QRS-axis as assessed by the ECG machine's algorithm as well as the intervals RR, PR, QRS and QT measured semi-automatically.

Heart rate (HR) and the QT interval corrected for HR (QTc e.g. QTcF and QTcB) will be determined by the sponsor (see TSAP for details).

All semi-automatic interval measurements in one subject will be performed on the same lead. The intervals will be measured from four cardiac cycles (beats) in lead II. If lead II shows a flat T wave or is not measurable for any reason, lead V5 will be used, or if that lead is not measurable, then lead I will be used. The lead actually used will be reported in the CTR.

For automatic interval measurements no lead will be provided.

For blinding arrangements see <u>section 4.1.5.1.</u> No more than two blinded readers will evaluate all ECGs of the study. ECGs from a particular subject should be evaluated by a single reader. For quality assurance and control of the measurements, all ECGs of a

c17703547-05  Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

subject will be subsequently reviewed by the ECG technician supervisor or his/her designee to assess the overall variance of the measured intervals and, to detect accidental switching of leads and/or false subject assignments of the ECGs. After quality control, the fiducial point markings will be reviewed by the cardiologist assigned to the study. Evaluation of ECGs will comply with the ICH E14 guidance document and supplements [R07-4722, R16-0366] as well as the FDA requirements for annotated digital ECGs [R09-4830].

#### b) Trial site

All local ECGs will be evaluated by the investigator or a designee.

For the inclusion or exclusion (see section 3.3) of a patient and for the assessment of cardiac safety during the study, the QT and QTc values generated by the ECG machines or their manual corrections by the investigators will be used. In doubtful cases, ECGs may be sent upfront for centralised evaluation (see below). In this case, these centrally measured results would overrule any other results obtained.

Abnormal findings, irrespective of whether they originate from central or local evaluation, will be reported as AEs (during the trial) or baseline conditions (at screening) if judged clinically relevant by the investigator. Any ECG abnormalities will be monitored carefully and, if necessary, the patient will be removed from the trial and will receive the appropriate medical treatment.

#### 5.2.5 Assessment of other safety parameters

#### 5.2.5.1 Vital signs

Systolic and diastolic BP as well as HR (considered to be equal to PR) will be measured by a blood pressure monitor at the times indicated in the Flow Chart, after patients have rested for at least 10 min in a supine position. All recordings should be made using the same type of blood pressure recording instrument on the same arm if possible. Further, respiratory rate [RR] and oral body temperature will be monitored. Body temperature will be determined at the time points indicated in the Flow Chart using electronic thermometers. Respiratory rate will be counted by trained study personal by observing the chest movements over a period of one minute after the subject has rested in the supine position for 5 minutes. Recording of the values will be done at the time points indicated in the Flow Chart.

#### 5.2.5.2 Medical examinations

At the screening visit, after informed consent is obtained, the medical examination will include documentation of patient information, demographics including height and body weight, smoking and alcohol history, relevant medical history and concomitant therapy, review of inclusion and exclusion criteria, review of vital signs (BP, PR, body temperature, respiratory rate), 12-lead ECG, laboratory tests including fecal occult blood and fecal calprotectin testing, suicidality assessment (C-SSRS) and, and a physical examination. At the end of treatment (EOT) examination, it will include review of vital signs, 12-lead ECG, laboratory tests, and a physical examination with determination of weight. Body weight should be measured with the patient wearing indoor clothing and no shoes. For each


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

individual patient, weight should be measured consistently in the morning or afternoon at all visits.

#### 5.2.5.3 Suicidal risk assessed by the C-SSRS

For the marketed PDE4-inhibitors apremilast [R17-1427];[R17-1539];[R17-1540] and roflumilast [R17-1542] an increased risk of suicidality has been described. Therefore prospective suicidality monitoring, will be performed throughout this trial using the Columbia Suicidal Severity Rating scale (C-SSRS).

C-SSRS results will be reported in terms of AEs as described in <u>Section 5.2.2.1</u>.

For additional details refer to appendix 10.1.

#### 5.3 OTHER

#### 5.4 APPROPRIATENESS OF MEASUREMENTS

All measurements performed during this trial are standard measurements and will be performed in order to monitor patients' safety and to determine PK and pharmacodynamics (PD) parameters in an appropriate way. The scheduled measurements will allow monitoring of changes in vital signs, standard laboratory values, and ECG parameters that might occur as a result of administration of trial medication. The safety assessments are standard, are accepted for evaluation of safety and tolerability of an orally administered drug, and are widely used in clinical trials. The PK parameters and measurements outlined in section 5.5


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

are generally used assessments of drug exposure.

# 5.5 DRUG CONCENTRATION MEASUREMENTS AND PHARMACOKINETICS

Date and clock time of drug administration and PK sampling will be recorded in the CRFs.

The actual sampling times will be used for determination of PK parameters.

PK sampling times and periods may be adapted during the trial based on information obtained during trial conduct (e.g. preliminary PK data) including addition of samples and visits as long as the total blood volume taken per patient does not exceed 400 mL. Such changes would be implemented via non-substantial CTP Amendments.

#### 5.5.1 Pharmacokinetic endpoints

The following PK parameters will be determined, if feasible:

#### 5.5.1.1 Secondary endpoints

BI 1015550

After the first dose (Day 1):

- AUC<sub> $\tau$ ,1</sub> (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval  $\tau$  after administration of the first dose)
- C<sub>max</sub> (maximum measured concentration of the analyte in plasma)

After the last dose (Day 14):

- AUC<sub> $\tau$ ,ss</sub> (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval  $\tau$ )
- $C_{max,ss}$  (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval  $\tau$ )


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5.5.2 Methods of sample collection

#### 5.5.2.1 Plasma sampling for pharmacokinetic analysis

For quantification of drug plasma concentrations of BI 1015550, BI 764333 , venous blood will be collected using a pre-labeled EDTA containing blood drawing tube at the times indicated in the <u>Flow Chart</u>. Blood will be withdrawn by means of either an indwelling venous catheter or by venipuncture with a metal needle.

A detailed description of sample collection and handling is provided in the Lab Manual in the ISF.

After completion of the trial the plasma samples may be used for further methodological investigations, e.g. for stability testing, assessment of metabolites. However, only data related to the analyte and/or its metabolite(s) including anti-drug antibodies (if applicable) will be generated by these additional investigations. The study samples will be discarded after completion of the additional investigations but not later than 5 years after the final study report has been signed.

Boehringer Ingelheim BI Trial No.: 1305-0012 c17703547-05

ringer Ingelheim 27 Mar 2019

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 5.5.3 Analytical determinations

# 5.5.3.1 Analytical determination of plasma concentrations

**Trial Protocol** 

BI 1015550 and BI 764333 concentrations in plasma will be determined by a validated high performance liquid chromatography with tandem mass spectrometry (HPLC-MS/MS) assay. The analysis will be performed under the responsibility of Drug Metabolism and Pharmacokinetics, Boehringer Ingelheim Pharma GmbH & Co. KG, Biberach, Germany at a suitable contract research organization (CRO).

As described in <u>section 4.1.5</u>, the bioanalyst will be unblinded during sample analysis.


Boehringer Ingelheim BI Trial No.: 1305-0012 c17703547-05

Trial Protocol


27 Mar 2019

Boehringer Ingelheim BI Trial No.: 1305-0012

c17703547-05

**Trial Protocol** 


27 Mar 2019

Boehringer Ingelheim BI Trial No.: 1305-0012 c17703547-05

Trial Protocol


27 Mar 2019

c17703547-05  Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **INVESTIGATIONAL PLAN 6.**

#### 6.1 VISIT SCHEDULE

Exact times of measurements outside the permitted time windows will be documented. The acceptable time windows for visits are given in the Flow Chart.

Study measurements and assessments scheduled to occur 'before' trial medication administration on Day 1 are to be performed and completed within a 2 h-period prior to the trial drug administration (including blank values for PK

The acceptable deviation on profile days (day 1, day 14) from the scheduled time is as follows: For the first 4h after trial drug administration: vital signs and ECG, -10min and for laboratory tests  $\pm$  30 min. After the first four hours after drug administration, vitals, ECG and laboratory tests  $\pm 30$  min.

Effort should be made to ensure that drug administration occurs at same time every day +/-30 min. On day 1 and 14 extra care should be made to maintain consistency with accurate documentation of actual time of administration.

If scheduled in the Flow Chart at the same time as a meal, blood sampling, vital signs and 12lead ECG recordings have to be done first. Furthermore, if several measurements including venepuncture are scheduled for the same time, venepuncture should be the last of the measurements due to its inconvenience to the patient and possible influence on physiological parameters.

For planned individual plasma concentration sampling times refer to the Flow Chart. While these nominal times should be adhered to as closely as possible, the actual sampling times will be recorded and used for determination of PK parameter.

If a patient misses an appointment, it will be rescheduled if possible. The relevance of measurements outside the permitted time windows will be assessed no later than at the Blinded Report Planning Meeting.

#### 6.2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS

#### 6.2.1 Screening and run-in period(s)

After having been informed about the trial, all patients will give their written informed consent in accordance with ICH-GCP and local legislation prior to enrolment in the study.

For information regarding laboratory tests (including drug and virus screening), ECG, vital signs, and physical examination, refer to sections 5.2.3 to section 5.2.5.

An historical HRCT can be used to determine eligibility, providing the scan was performed within the past 12 months prior to screening. If historical scan is not available, or an available scan fails to meet the required image acquisition specification, an HRCT may be performed after consent to determine eligibility. All HRCT scans will be sent to a central vendor for


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

review and confirmation of IPF diagnosis, prior to randomization. HRCT should not be repeated for eligibility if previous scan was taken within the past 3 months.

If required, the HRCT scan should be performed as close to screening date as possible, preferably once eligibility is confirmed based on other parameters, to avoid unnecessary scans for patients who are found ineligible based on other criteria. HRCT scans will be sent to a central reviewer for confirmation of IPF diagnosis. Confirmation of diagnosis must be available prior to visit 2.

Screening period may be extended for administrative reasons. Approval should be obtained from the sponsor who will also determine if any tests specified in the protocol must be repeated before the randomization visit.

#### **6.2.2** Treatment period

During the treatment period, patients will take trial medication twice daily.

At least one visit (visit 3), will be conducted inpatient; during which time patients will be kept under close medical surveillance. The patients will be allowed to leave the trial site only after formal assessment and confirmation of their fitness by the investigator or designee.

On all other study days, the study will be performed in an ambulatory fashion.

In addition to clinic visits, daily phone calls are required between study visits to assess and collect AE information and confirm compliance until day 14, with weekly phone calls between study visits thereafter until end of treatment.

#### Inpatient Visit 3: Day 1 and 2

Visit 3 will span at minimum, a two day period, day 1 and 2.

All patients must be admitted (inpatient) at the morning of day 1, and kept under close medical surveillance for at least 2 hours following evening drug administration on day 2. The patients will then be allowed to leave the trial site after formal assessment and confirmation of their fitness by the investigator or designee.

Each patient will receive the first dose of BI 1015550 or placebo the morning of Day 1 and the second dose the evening of day 1. Patients will take BI 1015550 (or placebo) twice daily (b.i.d) from Day 1 onwards. Trial medication will be taken orally. At clinic visits, trial medication will be taken under direct supervision of the investigator or designee. Details on treatments and procedures of administration are described in section 4.1.4.

Patients will be given a diary to record intake of study medication taken at home since the last clinic visit, during the treatment period. At each visit, the diary will be collected and reviewed for compliance and a new diary will be dispensed.

Visit 8: Day 14


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Study participants are required to be on site under medical surveillance for approximately 16 hours at day 14 to allow for required sampling and safety assessments as outlined in the Flow Chart. The patients are permitted to leave the trial site after formal assessment and confirmation of their fitness by the investigator or designee. As an alternative, the patient may be admitted or relocated to a nearby facility overnight. No additional testing is required during this period.

#### General:

For details on time points and procedures for collection of plasma samples for PK analysis, refer to Flow Chart and section 5.5.2.

The safety measurements performed during the treatment period are specified in <u>section 5.2.</u> of this protocol and in the Flow Chart. For details on time points for all other trial procedures, refer to the Flow Chart. AEs and concomitant therapy will be assessed continuously from screening until the end of trial examination.

#### End of Treatment Visit:

The EOT visit is required for all patients. The EOT visit is conducted when patients have concluded treatment with BI 1015550.

For patients who complete the full treatment period, this will be after 4 weeks of treatment, at visit 9.

For patients who prematurely discontinue trial medication, for any reason prior to 4 weeks, the abbreviated EOT visit should be completed as indicated in the <u>Flow Chart</u>, as soon as possible after stopping treatment.

#### 6.2.3 Follow-up period and end of trial

A follow up period of a minimum of 7 days (+3 days) will be required. All patients will complete an end of trial visit, including patients who discontinue treatment early. For AE assessment, laboratory tests, recording of ECG and vital signs, and physical examination during the end of trial period, see sections 5.2.2 to 5.2.5.

All abnormal values (including laboratory parameters) that are judged clinically relevant by the investigator will be monitored using the appropriate tests until a return to a medically acceptable level is achieved. Adverse events persisting after trial completion must be monitored until they have normalised or have been sufficiently characterised.

The end of the trial as a whole is defined by the 'last regular visit completed by last patient' or 'end date of the last open AE' or 'date of the last follow-up test' or 'date of an AE has been decided as sufficiently followed-up', whichever is latest.
c17703547-05  Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

#### 7.1 STATISTICAL DESIGN - MODEL

#### 7.1.1 **Objectives**

Trial objectives are given in Section 2.2.

The primary safety endpoint is defined in section 5.2.1. Inferential statistics are not planned (as explained in section 7.2).

PK endpoints as specified in section 5.5.1 will be analysed by descriptive statistics. Trough concentration values of BI 1015550 will be analysed regarding attainment of steady state as a pre-requisite for calculation of steady state parameters.

#### 7.2 NULL AND ALTERNATIVE HYPOTHESES

Safety and tolerability of different dose strengths of BI 1015550 are to be determined on the basis of the investigated parameters in comparison to placebo. It is not planned to test any statistical hypotheses with regard to these variables in a confirmatory sense. Instead, they will be described in their entirety and evaluated by descriptive statistical methods.

Confidence intervals will be computed and will have to be interpreted in the perspective of the exploratory character of the study, i.e. confidence intervals are considered as interval estimates for effects.

#### 7.3 PLANNED ANALYSES

All individual data will be listed.

Adherence to the protocol (such as inclusion/exclusion criteria, times of measurement, compliance with intake of trial medication, treatment dispensing errors, prohibited concomitant medication, completeness and consistency of data) will be checked. Important protocol deviations will be identified no later than in the Blinded Report Planning Meeting and provided in the TSAP.

#### 7.3.1 **Primary analyses**

Analysis of safety and tolerability is described in section 7.3.3.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.3.2 Secondary analyses

The secondary PK parameters (refer to <u>section 5.5.1</u>) will be calculated according to the BI SOP 'Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics' (01-MCS-36-472).

Plasma concentration data and parameters of a subject will be included in the statistical PK analyses if they are not flagged for exclusion due to a protocol violation relevant to the evaluation of PK (to be decided no later than in the Blinded Report Planning Meeting) or due to PK non-evaluability (as revealed during data analysis, based on the criteria specified below). Exclusion of a subject's data will be documented in the CTR.

Relevant protocol violations may be

- Incorrect trial medication taken, i.e. the subject received at least one dose of trial medication the subject was not assigned to
- Incorrect dose of trial medication taken
- Use of restricted medications.

Plasma concentrations and/or parameters of a subject will be considered as non-evaluable, if for example

- the subject experienced emesis that occurred at or before two times median t<sub>max</sub> of the respective treatment (Median t<sub>max</sub> is to be determined excluding the subjects experiencing emesis),
- missing samples/concentration data at important phases of PK disposition curve.

The PK parameter analysis set (PKS) includes all subjects in the Treated Set (TS) who provide at least one PK parameter that was not excluded according to the description above.

#### Attainment of steady state

Attainment of steady state will be explored by using the trough concentrations of BI 1015550 and BI 764333 between days 2 and 14 and the concentrations taken directly at the end of the dosing interval after the first drug administration and after the morning administration on Day 14 ( $C_{\tau,1}$ ,  $C_{\tau,27}$ ) for each dose level.

A nonlinear mixed effects model will be used to estimate the time to reach steady-state according to Hoffman et al. [R05-0788]. Accordingly, the observed trough plasma concentration  $C_{ij}$  for subject i after the  $j^{th}$  administration can be fitted by the following model:

$$C_{ij} = C_{ss} \cdot \exp(c_i) \cdot (1 - \exp(-(\gamma \cdot \exp(g_i) \cdot j))) \cdot \exp(e_{ij})$$

where

 $C_{ss}$  is the average steady-state trough concentration in the population,

 $c_i$  is the random deviation from  $C_{ss}$  with respect to subject i,

 $\gamma$  is the average first-order elimination rate in the population,


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- $g_i$  is the random deviation from  $\gamma$  with respect to subject i,
- $e_{ij}$  is the i.i.d. normally distributed random within-subject error ( $\sim N(0, \sigma_e^2)$ ).

The random effects  $c_i$  and  $g_i$  are multivariate normal distributed and independent of  $e_{ij}$ :

$$\begin{pmatrix} c_i \\ g_i \end{pmatrix} \sim N \left( \begin{pmatrix} 0 \\ 0 \end{pmatrix}, \begin{pmatrix} \sigma_c^2 & \sigma_{gc} \\ \sigma_{gc} & \sigma_g^2 \end{pmatrix} \right).$$

The time-point of sufficient approximation to the steady-state asymptote concentration is then determined from the fitted function. In other words, the time  $t_f$  to reach f = 85, 90 and 95% of steady-state can be calculated as follows:

$$t_f = \log(1 - f) / (-\gamma),$$

where  $\gamma$  is again the average first-order elimination rate in the population.

#### **Graphical displays**

To support the analyses of attainment of steady state, graphical representations of the data might be created. These might include (but are not limited to) individual time-courses of trough plasma concentrations and the (geometric) mean plasma concentration time profiles.

#### 7.3.3 Safety analyses

Safety will be assessed for the endpoints and parameters of interest listed in <u>section 5.2.1</u>. All treated patients (that is, all patients who received at least one dose of study drug), will be included in the safety evaluation. Safety analyses will be descriptive in nature and will be based on BI standards.

Treatments will be compared in a descriptive way. The placebo control group in the safety evaluation will consist of all placebo treated patients, regardless of the dose group in which they were treated. The active treatment groups will be compared to the placebo group in a descriptive way. Tabulations of frequencies/proportions will be used for the evaluation of categorical (qualitative) data, and tabulations of descriptive statistics will be used to analyse continuous (quantitative) data.

The analyses will be done by 'treatment at onset'.

Adverse events will be coded using the Medical Dictionary for Drug Regulatory Activities (MedDRA). Standard BI summary tables and listings will be produced. All adverse events with an onset between start of treatment and end of the residual effect period (REP), a period of 7 days after the last dose of trial medication, will be assigned to the on-treatment period for evaluation.

Statistical analysis and reporting of adverse events will concentrate on treatment-emergent adverse events, i.e. all adverse events occurring between start of treatment and end of the REP. Adverse events that start before first drug intake and deteriorate under treatment will also be considered as 'treatment-emergent'.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Frequency, severity, and causal relationship of adverse events will be tabulated by system organ class and preferred term after coding according to the current version of the MedDRA at the database lock.

Measurements (such as ECG, vital signs, or laboratory parameters) or AEs will be assigned to treatments (see <a href="section 4.1">section 4.1</a>) based on the actual treatment at the planned time of the measurement or on the recorded time of AE onset (concept of treatment emergent AEs). Therefore, measurements planned or AEs recorded prior to first intake of trial medication will be assigned to 'screening', those between first trial medication intake and end of REP will be assigned to the treatment period, and all AEs occurring between the end of REP and trial termination date will be assigned to 'follow-up'. These assignments including the corresponding time intervals will be defined in detail in the TSAP. Please note that AEs occurring after the last per protocol contact but entered before database lock will be reported to drug safety only and will not be captured in the trial database.

Additionally, further treatment intervals (analysing treatments) may be defined in order to provide summary statistics for time intervals, such as combined treatments, on-treatment totals or periods without treatment effects (such as screening and post-study intervals).

Laboratory data will be analysed both quantitatively as well as qualitatively. The latter will be done via comparison of laboratory data to their reference ranges. Values outside the reference range as well as values defined as clinically relevant will be summarised. Additionally, differences from baseline will be evaluated.

For vital signs, the differences from baseline will be evaluated.

The ECG variables QT, PR, QRS, and RR are obtained from the centralised evaluation of 12-lead ECG recordings.

The ECG variables HR, QTcF, QTcB will be derived from QT and RR interval obtained from central ECG evaluation.

These variables will be the basis for the derivation of quantitative and categorical ECG endpoints. The endpoints and their analyses will be described in the TSAP.

#### 7.3.4 Interim analyses

A preliminary analysis of PK parameters (AUC<sub>0-24</sub> and  $C_{max}$  of BI 1015550), provided as individual values and gMean of the first cohort per dose level, will be performed before proceeding to the next dose.

(Note: Data from the first cohorts of the above mentioned dose levels will be sufficient as long as the data from at least 4 patients on active drug were available)

In contrast to the final PK calculations, the preliminary analysis may be based on planned sampling times rather than on actual times, regardless of whether actual times were within the time windows or not. Therefore, minor deviations of preliminary and final results may occur. The preliminary analysis will provide individual and mean concentration/effect-time profiles and summary statistics of individual values without patient identification. The preliminary results will be distributed to the Investigator and the trial team.

**Trial Protocol** 


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Depending on the results of available preliminary PK analyses, the tolerability and safety of the compound, and changes of dosing schedule (e.g. additional intermediate doses) additional PK preliminary analysis may be performed based on the request of the clinical trial leader, the investigator, or Trial Clinical Pharmacokineticist. No formal preliminary PK/PD report will be written.

No formal inferential statistical interim analysis is planned. However, after each dose group, summaries and listings may be created to support the safety reviews. The investigator (or deputy) is allowed to postpone further dose progression until a preliminary analysis of the data already obtained has been performed

#### 7.3.5 Pharmacokinetic analyses

The PK parameters listed in <u>section 5.5.1</u> for drug BI 1015550 will be calculated according to the BI SOP 'Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics' (01-MCS-36-472).

Patients who are not included in the PKS (refer to <u>section 7.3.1</u>.) will be reported with their individual plasma concentrations and individual PK parameters; however, they will not be included in descriptive statistics for plasma concentrations, PK parameters or other statistical assessment.

Only concentration values within the validated concentration range and actual sampling times will be used for the calculation of PK parameters. Concentrations used in the PK calculations will be in the same format provided in the bioanalytical report, (that is, to the same number of decimal places provided in the bioanalytical report).


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.4 HANDLING OF MISSING DATA

## **7.4.1** Safety

c17703547-05

With respect to safety evaluations, it is not planned to impute missing values.

#### 7.4.2 Plasma drug concentration - time profiles

Handling of missing PK data will be performed according to the relevant SOP of the Sponsor (01-MCS-36-472).

Drug concentration data identified with no sample available (NOS), no valid result (NOR), not analysed (NOA), or below the lower limit of quantification (BLQ) will be displayed as such and not replaced by zero at any time point (this rule also applies to the lag phase, including the pre-dose values).

#### 7.4.3 Pharmacokinetic parameters

Handling of missing PK data will be performed according to the relevant SOP of the Sponsor (01-MCS-36-472).

For the non-compartmental analysis, concentration data identified with NOS, NOR or NOA will generally not be considered. Concentration values in the lag phase identified as BLQ will be set to zero. All other BLQ values of the profile will be ignored. The lag phase is defined as the period between time zero and the first time point with a concentration above the quantification limit.

#### 7.5 RANDOMISATION

Patients will be randomised within each dose/treatment group in a 2:1 ratio, which reflects the ratio of patients receiving active drug to placebo.

The sponsor will arrange for the randomisation as well as packaging and labelling of trial medication. The randomisation list will be generated using a validated system, which involves a pseudo-random number generator and a supplied seed number so that the resulting allocation is both reproducible and non-predictable.

The randomisation list will contain additional blocks to allow for patient replacement (refer to section 3.3.5).

#### 7.6 DETERMINATION OF SAMPLE SIZE

It is planned to include a total of 18 patients in this trial.

Additional patients may be entered to allow testing of additional intermediate doses within the planned dose range on the basis of experience gained during trial conduct (e.g. preliminary PK data), i.e. the actual number of patients entered may exceed 18.

**Trial Protocol** 


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The planned sample size is not based on a power calculation. The size of 9 patients per dose group (6 on active treatment, and 3 on placebo) is commonly used in multiple-rising dose studies of the present type and is in general considered as sufficient for the exploratory evaluation of multiple dose safety and PK.

An additional 6 patients (4 on active, 2 on placebo) will be entered in dose group 1A (18mg bid), therefore the total number of patients planned to be included in the trial is up to 24.

c17703547-05


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8. INFORMED CONSENT, DATA PROTECTION, TRIAL RECORDS

The trial will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, in accordance with the ICH-GCP and relevant BI SOPs.

The investigator should inform the sponsor immediately of any urgent safety measures taken to protect the study patients against any immediate hazard, and also of any serious breaches of the protocol or of ICH-GCP.

The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in a separate agreement between the investigator or the trial site and the sponsor. As a general rule, no trial results should be published prior to finalisation of the CTR.

# 8.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This trial will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB) / Independent Ethics Committee (IEC) and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

Prior to a patient's participation in the trial, written informed consent must be obtained from each patient (or the patient's legally accepted representative) according to ICH-GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional subject information form are to be retained by the investigator as part of the trial records. A copy of the signed and dated written informed consent and any additional subject information must be given to each patient or the patient's legally accepted representative.

The patient must be informed that his/her personal trial-related data will be used by Boehringer Ingelheim in accordance with the local data protection law. The level of disclosure must also be explained to the patient.

The patient must be informed that his or her medical records may be examined by authorised monitors CML/CRA or Clinical Quality Assurance auditors appointed by Boehringer Ingelheim, by appropriate IRB/IEC members, and by inspectors from regulatory authorities.

## 8.2 DATA QUALITY ASSURANCE

A quality assurance audit/inspection of this trial may be conducted by the sponsor or sponsor's designees, by IRBs/IECs, or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's trial-related files and correspondence, and the informed consent documentation of this clinical trial.

The data management procedures to ensure the quality of the data are described in detail in the trial data management and analysis plan (TDMAP) available in the clinical TMF.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8.3 RECORDS

c17703547-05

CRFs for individual patients will be provided by the sponsor. See <u>section 4.1.5.2</u> for rules about emergency code breaks. For drug accountability, refer to <u>section 4.1.8.</u>

#### **8.3.1** Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

All data reported in the CRFs must be consistent with the source data or the discrepancies must be explained.

The investigator may need to request previous medical records or transfer records, depending on the trial.

#### 8.3.2 Direct access to source data and documents

The investigator/institution will permit trial-related monitoring, audits, IRB/IEC review and regulatory inspection, providing direct access to all related source data/documents. CRFs and all source documents, including progress notes (if applicable) and copies of laboratory and medical test results must be available at all times for review by the sponsor's clinical trial monitor, auditor and inspection by health authorities (e.g. FDA). The CRA /on site monitor and auditor may review all CRFs, and written informed consents. The accuracy of the data will be verified by reviewing the documents described in section 8.3.1.

#### 8.4 LISTEDNESS AND EXPEDITED REPORTING OF ADVERSE EVENTS

#### 8.4.1 Listedness

To fulfil the regulatory requirements for expedited safety reporting, the sponsor evaluates whether a particular AE is 'listed', i.e. is a known side effect of the drug. Therefore a unique reference document for the evaluation of listedness needs to be provided. For BI 1015550 this is the current version of the Investigator's Brochure (c02094779-03). The current version of this reference document is to be provided in the ISF.

#### 8.4.2 Expedited reporting to health authorities and IECs/IRBs

Expedited reporting of SAEs, e.g. SUSARs to health authorities and IECs/IRBs, will be done according to local regulatory requirements. Further details regarding this reporting procedure are provided in the ISF.

#### 8.5 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this trial is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

Treatment data may be provided to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated as a result of the trial

Boehringer Ingelheim BI Trial No.: 1305-0012 c17703547-05

27 Mar 2019


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**Trial Protocol** 

need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB/IEC and the regulatory authorities, i.e. the CA.

#### 8.6 COMPLETION OF TRIAL

The EC/competent authority in each participating EU member state needs to be notified about the end of the trial (last patient/patient out, unless specified differently in <u>section 6.2.3</u> of the CTP) or early termination of the trial.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 9. REFERENCES

#### 9.1 PUBLISHED REFERENCES

| P05-12782 | Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, Grinten CPM van der, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J. Standardisation of spirometry. Eur Respir J 26 (2), 319 - 338 (2005). |
|---|---|
| P06-08316 | Giembycz MA. An update and appraisal of the cilomilast phase III clinical development programme for chronic obstructive pulmonary disease. Br J Clin Pharmacol 2006;62(2):138-152. |
| P11-07084 | Raghu G, et al, ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med 2011;183(6):788-824. |
| P15-07539 | Raghu G, et al, American Thoracic Society (ATS), European Respiratory Society (ERS), Japanese Respiratory Society (JRS), Latin American Thoracic Association (ALAT). An official ATS/ERS/JRS/ALAT clinical practice guideline: treatment of idiopathic pulmonary fibrosis: an update of the 2011 clinical practice guideline. Am J Respir Crit Care Med 2015;192(2):e3-e19. |
| R05-0788 | Hoffman D, Kringle R, Lockwood G, Turpault S, Yow E, Mathieu G. Nonlinear mixed effects modelling for estimation of steady state attainment. Pharm Stat 4, 15 - 24 (2005). |
| R06-2002 | Macintyre N, Crapo RO, Viegi G, Johnson DC, Grinten CPM van der, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, Gustafsson P, Hankinson J, Jensen R, McKay R, Miller MR, Navajas D, Pedersen OF, Pellegrino R, Wanger J. Standardisation of the single-breath determination of carbon monoxide uptake in the lung. Eur Respir J 2005; 26:720-35. |
| R07-4722 | Guidance for industry: E14 clinical evaluation of QT/QTc interval prolongation and proarrhythmic potential for non-antiarrhythmic drugs. Rockville: U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), Center for Biologics Evaluation and Research (CBER) (2005) |
| R09-4830 | Brown BD, Badilini F. HL7 aECG implementation guide (March 21, 2005). |

| R10-1555 | Daxas (roflumilast) in chronic obstructive pulmonary disease, NDA 22-522, FDA Advisory Committee briefing document presented to: Pulmonary-Allergy Drugs Advisory Committee (briefing book, April 7, 2010). website.fda.gov/AdvisoryCommittees/CommitteesMeetingMaterials/Drugs/Pulmonary-AllergyDrugsAdvisoryCommittee/ucm207376.htm (access date: 23 November 2010); Jersey City: Forest Research Institute; 2010. |
|---|---|
| R10-1559 | Giembycz MA. Life after PDE4: overcoming adverse events with dual-specificity phosphodiesterase inhibitors. Curr Opin Pharmacol 2005;5:238-244. |
| R11-2587 | Ley B, Collard HR, King TE. Clinical course and prediction of survival in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med 2011;183:431-440. |
| R12-5527 | Nalysnyk L, Cid-Ruzafa J, Rotella P, Esser D. Incidence and prevalence of idiopathic pulmonary fibrosis: review of the literature. Eur Respir Rev 2012; 21(126):355-361. |
| R14-1795 | Otezla (apremilast) tablets, for oral use (Celgene) (U.S. prescribing information, revised: 3/2014). |
| R16-0366 | E14 Implementation Working Group ICH E14 guideline: the clinical evaluation of QT/QTc interval prolongation and proarrhythmic potential for non-antiarrhythmic drugs: questions & answers (R3) (current version dated 10 December 2015). http://www.ich.org/fileadmin/Public_Web_Site/ICH_Products/Guidelines/E fficacy/E1 4/E14_Q_As_R3Step4.pdf (access date: 29 January 2015); Geneva: International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (2015) |
| R16-1924 | Gisbert JP, Bermejo F, Perez-Calle JL, Taxonera C, Vera I, McNicholl AG, Algaba A, Lopez P, Lopez-Palacinos N, Calvo M, Gonzalez-Lama Y, Cameros JA, Velasco M, Mate J. Fecal calprotectin and lactoferrin for the prediction of inflammatory bowel disease relapse. Inflamm Bowel Dis. 15 (8), 1190-1198 (2009). |
| R17-0158 | Korkmaz S, Maupoil V, Sobry C, et al. An increased regional blood flow precedes mesenteric inflammation in rats treated by a phosphodiesterase 4 inhibitor. Tox Sci 2009; 107(1):298-305. |
| R17-0915 | Roflumilast 500 mcg tablets (Forest Research Institute): pharmacology/toxicology NDA/BLA review and evaluation, application number: 022522Orig1s000. website.accessdata.fda.gov/drugsatfda_docs/nda/2011/022522Orig1s000Ph armR.pdf (access date: 13 March 2017); Department of Health and Human Services, Public Health Service, Food and Drug Administration, Center for Drug Evaluation and Research (2011) |

| R17-0916 | Losco PE, Evans EE, Barat SA, et al. The toxicity of SCH 351591, a novel |
|---|---|
| | phosphodiesterase-4 inhibitor, in cynomolgus monkeys. Toxicol Pathol |
| | 2004: 32:295-308. |

- R17-0919 Otezla (apremilast) (Celgene): pharmacology/toxicology NDA/BLA review and evaluation, application number: 205437Orig1s000. website.accessdata.fda.gov/drugsatfda docs/nda/2014/205437Orig1s000Ph armR.pdf (access date: 13 March 2017); Department of Health and Human Services, Public Health Service, Food and Drug Administration, Center for Drug Evaluation and Research (2014)
- R17-1427 Otezla 10 mg, 20 mg, 30 mg film-coated tablets, Otezla 30 mg film-coated tablets (Celgene) (summary for product characteristics, manufacturer responsible for batch release, conditions or restrictions regarding supply and use, other conditions and requirements of the marketing authorisation, conditions or restrictions with regard to the safe and effective use of the medicinal product, labelling and package leaflet (first published 16/02/2015). website.ec.europa.eu/health/documents/communityregister/2015/20 150115130395/anx 130395 en.pdf (access date: 19 April 2017); 2015.
- Otezla 30mg tablets (Celgene) (summary of product characteristics updated R17-1539 05-Jan-2017). website.medicines.org.uk/emc/printdocument?documentId=29792 (access date: 2 May 2017); 2017.
- R17-1540 Otezla 10mg, 20mg, 30mg treatment initiation pack (Celgene) (summary of product characteristics updated 05-Jan-2017). website.medicines.org.uk/emc/print-document?documentId=29793 (access date: 2 May 2017); 2017.
- R17-1542 Daxas 500 micrograms film-coated tablets (AstraZeneca) (summary of product characteristics updated 06-Dec-2016). website.medicines.org.uk/emc/print-document?documentId=23416 (access date: 2 May 2017); 2016.
- Graham BL, Brusasco V, Burgos F, et al. 2017 ERS/ATS standards for R17-3686 single-breath carbon monoxide uptake in the lung. Eur Respir J 2017; 49: 1600016 [https://doi.org/10.1183/13993003.00016-2016].

#### 9.2 UNPUBLISHED REFERENCES

- 01-MCS-36-472 Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics. Current version
- 001-MCG-312 Biomarker Assessments on Trial Level. Current version
- U10-3777-01 Investigator Brochure BI 137882 BS. 11 Feb 2011

c17703547-05

**Trial Protocol** 


| U13-1792-01 | Safety, tolerability and pharmacokinetics of single rising oral doses of BI 1015550 in healthy male volunteers (a partially randomised, single-blinded, placebo-controlled Phase I study). 1305.1. 21 Jun 2013 |
|---|---|
| c02094779-03 | Investigator's Brochure BI 1015550 for Idiopathic Pulmonary Fibrosis. 22Feb2018 |
| c02191718-02 | Safety, tolerability and pharmacokinetics of multiple rising oral doses of BI 1015550 powder for oral solution in healthy male volunteers q.d. or b.i.d. for 14 days (a randomised, double-blind, placebo-controlled within dose groups Phase I trial). 1305.2. 15 Apr 2014 |
| c20307414-01 | Final Clinical Trial Report (1305-0020). Relative bioavailability of BI 1015550 following oral administration under fed and fasted conditions in healthy male subjects. 16 July 2018 |
| c22991937-01 | Final Clinical Trial Report (1305-0011). Safety, tolerability, and pharmacokinetics of single (Part 1) and multiple rising oral doses (Part 2) of BI 1015550 in healthy male subjects. 15 November 2018 |

c17703547-05

Trial Protocol


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10. APPENDICES

### 10.1 COLUMBIA SUICIDAL SEVERITY RATING SCALE (C-SSRS)

The C-SSRS is a brief measure which is designed to assess severity and change of suicidality by integrating both, behavior and ideation. The C-SSRS was designed to address the need for a summary measure to track change in the severity of suicidality across both clinical settings and treatment trials.

At screening, C-SSRS (screening version) will be assessed with the aim to exclude patients with suicidal ideation type 2-5 within the preceding 12 months and patients with any lifetime history of suicidal behavior. Subsequently, the C-SSRS "since last visit" assessment will be performed at the time points given in the <u>Flow Chart.</u> For assessment, paper forms will be used and results will be transcribed into the CRF.

All positive reports during trial treatment are treatment-emergent adverse events (AEs). The results of further medical, including psychiatric examinations should be documented as adverse events where appropriate.

The original Columbia Suicidal Severity Rating scales used in this trial are shown as follows: Visit 1 –Screening version
Subsequent visits- Since last visit version.

c17703547-05 Trial Protocol 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Screening

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <a href="The Columbia Suicide History">The Columbia Suicide History</a>
Form, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc.

c17703547-05


| SUICIDAL IDEATION | | | |
|---|---|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suicidal Behavior" section. If the answer to question 2 is "yes", ask questions 3, 4 and 5. If the answer to question 1 and/or 2 is "yes", complete "Intensity of Ideation" section below. | | | Past<br>X Months |
| <ol> <li>Wish to be Dead Subject endorses thoughts about a wish to be dead or not alive anymore, or wish to fall asleep and not wake up. Have you wished you were dead or wished you could go to sleep and not wake up? </li> </ol> | | | No |
| If yes, describe: | | | |
| <ol> <li>Non-Specific Active Suicidal Thoughts General, non-specific thoughts of wanting to end one's life/commit suiconeself/associated methods, intent, or plan. Have you actually had any thoughts of killing yourself?</li> </ol> | tide (e.g., "T've thought about killing myzelf") without thoughts of ways to kill | Yes | No |
| If yes, describe: | | | |
| | thod during the assessment period. This is different than a specific plan with time, but not a specific plan). Includes person who would say, "I thought about taking an | Yes | No |
| If yes, describe: | | | |
| 4. Active Suicidal Ideation with Some Intent to Act, with Active suicidal thoughts of killing oneself and subject reports having as definitely will not do anything about them.— Have you had these thoughts and had some intention of acting on the | sme intent to act on such thoughts, as opposed to "I have the thoughts but I | Yes | No |
| If yes, describe: | | | |
| <ol> <li>Active Suicidal Ideation with Specific Plan and Intent<br/>Thoughts of killing oneself with details of plan fully or partially worked<br/>Have you started to work out or worked out the details of how to kill y</li> </ol> | d out and subject has some intent to carry it out. | Yes | No |
| If yes, describe: | | | |
| INTENSITY OF IDEATION | | | |
| The following features should be rated with respect to the most and 3 being the most severe). Ask about time heishe was feeling | zevere type of ideation (i.e., 1-5 from above, with 1 being the least severe the most suicidal. | М | ost |
| Most Severe Ideation: | | | vere |
| Type # (1-5) | Description of Ideation | | |
| Frequency How many times have you had these thoughts? (1) Less than once a week (2) Once a week (3) 2-5 times in w | eek (4) Daily or almost daily (5) Many times each day | - | _ |
| Duration When you have the thoughts, how long do they last? | | | |
| (1) Fleeting - few seconds or minutes (2) Less than 1 hour/some of the time (3) 1-4 hours/a lot of time (4) 4-8 hours/most of day (5) More than 8 hours/persistent or continuous | | | |
| Controllability Could/can you stop thinking about killing yourself or wanting to die if you want to? (1) Easily able to control thoughts (4) Can control thoughts with a lot of difficulty (5) Unable to control thoughts with some difficulty (0) Does not attempt to control thoughts | | | - |
| Deterrents Are there things - anyone or anything (e.g., family, religion, pain of death) - that stopped you from wanting to die or acting on thoughts of committing suicide? (1) Deterrents definitely stopped you from attempting suicide (2) Deterrents probably stopped you (3) Deterrents definitely did not stop you (5) Deterrents definitely did not stop you | | | _ |
| (3) Uncertain that deterrents stopped you | (0) Does not apply | | |
| | ing to die or killing yourself? Was it to end the pain or stop the way with this pain or how you were feeling) or was it to get attention, (4) Mostly to end or stop the pain (you couldn't go on living with the pain or how you were feeling) (5) Completely to end or stop the pain (you couldn't go on | _ | |
| and to end/stop the pain | living with the pain or how you were feeling) (0) Does not apply | Vest | - 1/1//00 |


| SUICIDAL BEHAVIOR (Check all that apply, 20 long as these are separate events; must ask about all types) | | | Past X Years<br>or<br>Lifetime |
|---|---|---|---|
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, as a result of act. Behavior was in part thought of as method to kill oneself. Intent does not have to be 100%. If there is any intent/desire to die associated with the act, then it can be considered an actual suicide attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger while gun is in mouth but gun is broken so no injury results, | | | Yes No |
| this is considered an attempt. Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumsta act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from window someone denies intent to die, but they thought that what they did could be lethal, intent may be inferred. | | | |
| Have you made a suicide attempt? Have you done anything to harm yourself? Have you done anything dangerous where you could have died? What did you do? | | | Total # of<br>Attempts |
| Did you as a way to end your life? Did you want to die (even a little) when you? Were you trying to end your life when you? Or did you think it was possible you could have died from? | | | _ |
| Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve str<br>or get something else to happen)? (Self-Injurious Behavior without suicidal intent)<br>If yes, describe: | ress, feel better | r, get sympathy, | |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? | | | Yes No |
| Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, a occurred). Overdoos: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rathe | r than an interrup | ted attempt. | Yes No |
| Shooting: Person has gan pointed toward self, gun is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so. Has there been a time when you started to do something to end your life but someone or something stopped you before you | | | Total # of interrupted |
| actually did anything? If yes, describe: | | | <u> </u> |
| Aborted Attempt: When person begins to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. Has there been a time when you started to do something to try to end your life but you stopped yourself before you actually did anything? If yes, describe: | | | Yes No |
| Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: | | | Yes No |
| Suicidal Behavior: Suicidal behavior was present during the assessment period? | | | Yes No |
| Answer for Actual Attempts Only Most Re Attempt Date | | Attempt | Initial/First<br>Attempt<br>Date: |
| Actual Lethality/Medical Damage: No physical damage or very minor physical damage (e.g., surface scratches). Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding; sprains). Modernte physical damage; medical amenton needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes intact; third-degree burns less than 20% of body, extensive blood loss but can recover; major fractures). Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body, extensive blood loss with unstable vital signs; major damage to a vital area). Death | | Enter Code | Enter Code |
| Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: pur gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). | Enter Code | Enter Code | Enter Code |
| 0 = Behavior not likely to result in injury 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death despite available medical care | _ | — | _ |

Trial Protocol


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# COLUMBIA-SUICIDE SEVERITY RATING SCALE (C-SSRS)

Since Last Visit

Version 1/14/09

Posner, K.; Brent, D.; Lucas, C.; Gould, M.; Stanley, B.; Brown, G.; Fisher, P.; Zelazny, J.; Burke, A.; Oquendo, M.; Mann, J.

#### Disclaimer:

This scale is intended to be used by individuals who have received training in its administration. The questions contained in the Columbia-Suicide Severity Rating Scale are suggested probes. Ultimately, the determination of the presence of suicidal ideation or behavior depends on the judgment of the individual administering the scale.

Definitions of behavioral suicidal events in this scale are based on those used in <u>The Columbia Suicide History</u> <u>Form</u>, developed by John Mann, MD and Maria Oquendo, MD, Conte Center for the Neuroscience of Mental Disorders (CCNMD), New York State Psychiatric Institute, 1051 Riverside Drive, New York, NY, 10032. (Oquendo M. A., Halberstam B. & Mann J. J., Risk factors for suicidal behavior: utility and limitations of research instruments. In M.B. First [Ed.] Standardized Evaluation in Clinical Practice, pp. 103-130, 2003.)

For reprints of the C-SSRS contact Kelly Posner, Ph.D., New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, 10032; inquiries and training requirements contact posnerk@nyspi.columbia.edu

© 2008 The Research Foundation for Mental Hygiene, Inc.


Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| SUICIDAL IDEATION | | | |
|---|---|---|---|
| Ask questions 1 and 2. If both are negative, proceed to "Suicidal Behavior" section. If the answer to question 2 is "yes", ask questions 3, 4 and 5. If the answer to question 1 and/or 2 is "yes", complete "Intensity of Ideation" section below. | | | |
| 1. With to be Dead | | Yes | w. |
| Subject endorses thoughts about a wish to be dead or not alive anymore, or wish to fall asleep and not wake up. Have you wished you were dead or wished you could go to sleep and not wake up? | | | No |
| If yes, describe: | | | |
| 2. Non-Specific Active Suicidal Thoughts | | | |
| General, non-specific thoughts of wanting to end one's life/commit suic | ide (e.g., "I've thought about killing myself") without thoughts of ways to kill | Yes | No |
| oneself'associated methods, intent, or plan during the assessment period<br>Have you actually had any thoughts of killing yourself? | | | |
| If yes, describe: | 200 to 100 to | 1.0 | |
| 3. Active Suicidal Ideation with Any Methods (Not Plan) | | Yes | No |
| place or method details worked out (e.g., thought of method to kill self) | thod during the assessment period. This is different than a specific plan with time, but not a specific plan). Includes person who would say, "I thought about taking an | | |
| overdose but I never made a specific plan as to when, where or how I w<br>Have you been thinking about how you might do this? | ould actually do itand I would never go through with it." | П | П |
| If yes, describe: | | | |
| 4. Active Suicidal Ideation with Some Intent to Act, with | nout Specific Plan | | |
| Active suicidal thoughts of killing oneself and subject reports having so<br>definitely will not do anything about them." | ome intent to act on such thoughts, as opposed to "I have the thoughts but $I$ | Yes | No |
| Have you had these thoughts and had some intention of acting on the | m? | | |
| If yes, describe: | | | |
| 5. Active Suicidal Ideation with Specific Plan and Intent | | | |
| Thoughts of killing oneself with details of plan fully or partially worked<br>Have you started to work out or worked out the details of how to kill y | | Yes | No |
| If yes, describe: | 1000 | | |
| INTENSITY OF IDEATION | | | |
| | severe type of ideation (i.e., 1-5 from above, with 1 being the least severe | | |
| and 5 being the most severe). | | l M | ost |
| Most Severe Ideation: | | | vere |
| Type # (1-5) | Description of Ideation | | |
| Frequency How many times have you had these thoughts? | American Company of the Company of t | | |
| (1) Less than once a week (2) Once a week (3) 2-5 times in we | eek (4) Daily or almost daily (5) Many times each day | _ | |
| Duration | | | |
| When you have the thoughts, how long do they last? (1) Fleeting - few seconds or minutes | (4) 4-8 hours/most of day | | _ |
| (2) Less than 1 hour/some of the time<br>(3) 1-4 hours/a lot of time | (5) More than S hours/persistent or continuous | | |
| Controllability | 0 | | |
| Could/can you stop thinking about killing yourself or want | ting to die if you want to? (4) Can control thoughts with a lot of difficulty | | |
| (1) Easily able to control thoughts (2) Can control thoughts with little difficulty | (5) Unable to control thoughts | - | _ |
| (3) Can control thoughts with some difficulty | (0) Does not attempt to control thoughts | _ | |
| Deterrents Are there things - anyone or anything (e.g., family, religior | n, pain of death) - that stopped you from wanting to die or acting on | | |
| thoughts of committing suicide? | (A) T. (B) A. (B | | |
| <ol> <li>Deterrents definitely stopped you from attempting suicide</li> <li>Deterrents probably stopped you</li> </ol> | (4) Deterrents most likely did not stop you<br>(5) Deterrents definitely did not stop you | _ | |
| (3) Uncertain that deterrents stopped you | (0) Does not apply | _ | |
| | | 1 | |
| Reasons for Ideation What sort of reasons did you have for thinking about want | ing to die or killing yoursel? Was it to end the pain or you the way | 1 | |
| What sort of reasons did you have for thinking about want<br>you were feeling (in other words you couldn't go on living | ing to die or killing yourself? Was it to end the pain or stop the way with this pain or how you were feeling) or was it to get attention, | | |
| What sort of reasons did you have for thinking about want | | | _ |
| What sort of reasons did you have for thinking about wants<br>you were feeling (in other words you couldn't go on living<br>revenge or a reaction from others? Or both?<br>(1) Completely to get attention, revenge or a reaction from others<br>(2) Mostly to get attention, revenge or a reaction from others | with this pain or how you were feeling) or was it to get attention, (4) Mostly to end or stop the pain (you couldn't go on living with the pain or how you were feeling) | _ | _ |
| What sort of reasons did you have for thinking about want,<br>you were feeling (in other words you couldn't go on living<br>revenge or a reaction from others? Or both?<br>(1) Completely to get attention, revenge or a reaction from others | with this pain or how you were feeling) or was it to get attention, (4) Mostly to end or stop the pain (you couldn't go on | - | |

Version 1/14/0


| SUICIDAL BEHAVIOR (Check all that apply, so long as these are separate events; must ask about all types) | Since Last<br>Visit |
|---|---|
| Actual Attempt: A potentially self-injurious act committed with at least some wish to die, at a result of act. Behavior was in part thought of as method to kill oneself. Intent does not have to be 100%. If there is any intentidesize to die associated with the act, then it can be considered an actual suicide attempt. There does not have to be any injury or harm, just the potential for injury or harm. If person pulls trigger while gan is in mouth but gan is broken so no injury results, this is considered an attempt. Inferring Intent: Even if an individual denies intent/wish to die, it may be inferred clinically from the behavior or circumstances. For example, a highly lethal act that is clearly not an accident so no other intent but suicide can be inferred (e.g., gunshot to head, jumping from window of a high floor/story). Also, if someone denies intent to die, but they thought that what they did could be lethal, intent may be inferred. Have you made a suicide attempt? Have you more anything to harm yourself? | Yes No |
| Have you done anything dangerous where you could have died? What did you do? Did you as a way to end your life? Did you want to die (even a little) when you? Were you trying to end your life when you? Or did you think it was possible you could have died from? Or did you do it purely for other reasons / without ANY intention of killing yourself (like to relieve stress, feel better, get sympathy, or get something else to happen)? (Self-Injurious Behavior without suicidal intent) If yes, describe: | Total # of<br>Attempts |
| | Yes No |
| Has subject engaged in Non-Suicidal Self-Injurious Behavior? Interrupted Attempt: When the person is interrupted (by an outside circumstance) from starting the potentially self-injurious act (if not for that, actual attempt would have occurred). Overdose: Person has pills in hand but is stopped from ingesting. Once they ingest any pills, this becomes an attempt rather than an interrupted attempt. Shooting: Person has gun pointed toward self, gun is taken away by someone else, or is somehow prevented from pulling trigger. Once they pull the trigger, even if the gun fails to fire, it is an attempt. Jumping: Person is poised to jump, is grabbed and taken down from ledge. Hanging: Person has noose around neck but has not yet started to hang - is stopped from doing so. Has there been a time when you started to do something to end your life but someone or something stopped you before you actually did anything? | Yes No |
| If yes, describe: | _ |
| Aborted Attempt: When person begans to take steps toward making a suicide attempt, but stops themselves before they actually have engaged in any self-destructive behavior. Examples are similar to interrupted attempts, except that the individual stops him/herself, instead of being stopped by something else. Has there been a time when you started to do something to try to end your life but you stopped yourself before you actually did anything? If yes, describe: | Yes No Total # of aborted |
| Preparatory Acts or Behavior: Acts or preparation towards imminently making a suicide attempt. This can include anything beyond a verbalization or thought, such as assembling a specific method (e.g., buying pills, purchasing a gun) or preparing for one's death by suicide (e.g., giving things away, writing a suicide note). Have you taken any steps towards making a suicide attempt or preparing to kill yourself (such as collecting pills, getting a gun, giving valuables away or writing a suicide note)? If yes, describe: | Yes No |
| Suicidal Behavior: Suicidal behavior was present during the assessment period? | Yes No |
| Suicide: | Ves No |
| Answer for Actual Attempts Only | Most Lethal Attempt Date: |
| Actual Lethality/Medical Damage: 0. No physical damage or very minor physical damage (e.g., surface scratches). 1. Minor physical damage (e.g., lethargic speech; first-degree burns; mild bleeding, sprains). 2. Moderate physical damage, medical amention needed (e.g., conscious but sleepy, somewhat responsive; second-degree burns; bleeding of major vessel). 3. Moderately severe physical damage; medical hospitalization and likely intensive care required (e.g., comatose with reflexes innect; third-degree burns less than 20% of body; extensive blood loss but can recover, major fractures). 4. Severe physical damage; medical hospitalization with intensive care required (e.g., comatose without reflexes; third-degree burns over 20% of body; extensive blood loss with unstable vital signs; major damage to a vital area). 5. Death | Enter Code |
| Potential Lethality: Only Answer if Actual Lethality=0 Likely lethality of actual attempt if no medical damage (the following examples, while having no actual medical damage, had potential for very serious lethality: put gun in mouth and pulled the trigger but gun fails to fire so no medical damage; laying on train tracks with oncoming train but pulled away before run over). 0 = Behavior not likely to result in injury | Enter Code |
| 1 = Behavior likely to result in injury but not likely to cause death 2 = Behavior likely to result in death demits available medical care | _ |

Boehringer Ingelheim BI Trial No.: 1305-0012

c17703547-05

**Trial Protocol** 


27 Mar 2019

#### **DESCRIPTION OF GLOBAL AMENDMENT(S)** 11.

| Number of global amendment | 1.0 |
|---|---|
| Date of CTP revision | 21 Jun 2018 |
| EudraCT number | 2017-002736-16 |
| BI Trial number | 1305-0012 |
| BI Investigational Product(s) | BI 1015550 |
| Title of protocol | Safety, tolerability, and pharmacokinetics of |
| | multiple rising oral doses of BI 1015550 in patients with idiopathic pulmonary fibrosis (IPF) on no background anti-fibrotic (Part 1) and safety and tolerability of BI 1015550 on top of Nintedanib and Pirfenidone (Part 2) |
| To be implemented as the | |
| To be implemented only after | |
| approval of the IRB / IEC / | |
| Competent Authorities | |
| To be implemented | |
| immediately in order to eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | |
| IRB / IEC / Competent | |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | |
| , v | |
| Section to be changed | Flow chart 1A- MRD Overview |
| | Flow chart 1B- part 1: Visit 3 |
| | Flow chart 1C- part 1: Visit 8 |
| Description of change | |
| Rationale for change | The risk of human disproportionate metabolite is |
| | turned out to be low based on the recently |
| | available metabolite identification data from |
| | Study 1305-0011. Therefore, samplings for |


| Number of global amendment | 1.0 |
|---|---|
| Number of global amenument | metabolite identification were eliminated to |
| | reduce the burden of patients. |
| Coation to be abouted | Elevy about 2A COC Oversions |
| Section to be changed | Flow chart 2A: SOC Overview |
| Description of change | Phone visit: |
| | Compliance check removed from part 2 flow |
| | chart |
| | Concomitant therapy added to part 2 flow chart |
| Rationale for change | Phone visits updated for consistency between |
| | part1 and 2 |
| Section to be changed | Flow chart 1A: MRD Overview |
| | Flow chart 2A: SOC Overview |
| Description of change | Footnote 13 regarding pre dose PK samples, |
| | updated for clarification that day 84 (part 1) and |
| | day 28 (part 2) pk samples are taken the morning |
| | of the visit, similar to other samples listed. These |
| | samples are not considered pre dose as there is no |
| | dosing at day 84 (part 1) or day 28 (part 2) and |
| | are therefore considered post (previous day) dose. |
| Rationale for change | Clarification |
| Section to be changed | Abbreviations |
| Description of change | Columbia-suicide severity ranking score corrected |
| | to Columbia-suicide severity rating scale |
| Rationale for change | Correction |
| | · |
| Section to be changed | 1.2.4 |
| Description of change | Missing information about CYP3A induction and |
| | no clinically relevant PK-DDI potential of BI |
| | 1015550 with nintedanib and pirfenidone was |
| | added. |
| Rationale for change | Updated as applicable to DDI potential with SOC. |
| 0 | 1 1 |
| Section to be changed | 1.2.5.1.3 |
| | 1.2.5.2.2 |
| <b>Description of change</b> | Preliminary results pertaining to clinical safety |
| 1 | and clinical pharmacokinetics for trial 1305-0011 |
| | added to introduction section. |
| Rationale for change | Preliminary results have become available since |
| | finalization of protocol. |
| <u> </u> | |
| Section to be changed | 1.2.5.1.4 |
| bection to be changed | 1.2.5.2.3 (new section added) |
| | 1.2.3.2.3 (new section added) |


| Number of global amendment | 1.0 |
|---|---|
| Description of change | Preliminary results pertaining to clinical safety and clinical pharmacokinetics for trial 1305-0020 added to introduction section. |
| Rationale for change | Preliminary results have become available since finalization of protocol |
| Section to be changed | 1.2.5.2.3 updated to section 1.2.5.2.4 |
| Description of change | Statement "Exposure estimate will be updated to |
| | include PK data from ongoing trials (1305.11, 1305.20) as they become available" has been removed and the respective expected exposures in Section 1.2.5.2.4 were updated. |
| Rationale for change | PK information has been updated and therefore statement is no longer applicable. |
| Section to be changed | 3.1.1 |
| Description of change | Additional description added regarding meeting with investigators |
| Rationale for change | This will ensure key findings of safety review committee are outlined with investigators and investigators have intimate knowledge of the data. |
| Section to be changed | 3.3 |
| Description of change | Description of re-screening added. |
| Rationale for change | Re-screening may be permitted in specific circumstances. Clarification in protocol added to ensure sites are aware of requirements. |
| Section to be changed | 3.3.3 |
| Description of change | Exclusion 3, cholecystectomy removed. |
| Rationale for change | Cholecystectomy was eliminated from the exclusion criteria because food effect trial show negligible effect of food on AUC and the risk that cholecystectomy could interfere with PK of BI 1015550 is low considering the contribution of major drug transporters in BI 1015550 disposition is minimal based on in vitro data. |
| Section to be shanged | 3.3.3 |
| Description of change | Exclusion 17 updated with respect to abstinence requirements. |
| Rationale for change | Clarification that only true abstinence is Permitted. Periodic abstinence (e.g calendar, ovulation), declaration of abstinence for the duration of exposure to IMP, and withdrawal are |

| Number of global amendment | 1.0 |
|---|---|
| | not acceptable methods of contraception |
| | • |
| Section to be changed | 3.3.3 and table 4.2.2.1:1 |
| Description of change | Exclusion 20 updated- prior use of SOC is |
| I am I am B | acceptable, but restricted if taken within 30 days |
| | prior to screening (V1). |
| Rationale for change | More in line with clinical practice. Patients are |
| | often tried on antifibrotic therapy for longer than |
| | 3 months before discontinuation due to the |
| | severity of the disease. Time window of 30 days |
| | is considered adequate to minimize any potential |
| | carried over effects of these treatments on the PK |
| | and safety of BI 1015550. |
| Section to be changed | 4.1.3.1 |
| Description of change | Table 4.1.3.1 was updated based on the most |
| | recent data. |
| Rationale for change | Expected exposure in the present trial in Table |
| _ | 4.1.3.1 was updated based on the most recent data |
| | (1305-0011 and 1305-0020). |
| _ | |
| Section to be changed | 4.2.2.1 |
| Description of change | Clarification to medication restrictions part 2 |
| | Table 4.2.2.1:2, footnote 7 added, additional text |
| | in note |
| Rationale for change | Clarifications of potential drug-drug interactions |
| | as applicable to pirfenidone SOC. |
| Section to be changed | 5.2.3 |
| Description of change | Clarification that stool sample collection 3 days |
| | prior to first dose is collected as v2 (day (-1) |
| | sample. No sample is required at randomization |
| D.C. L.C. L | (day 1). |
| Rationale for change | Correction |
| | 500 m 11 5000 i |
| Section to be changed | 5.2.3 Table 5.2.3:1 |
| Description of change | Glutamate dehydrogenase (GLDH) removed as a |
| | required parameter to be measured. |
| Rationale for change | Based on current liver safety profile collected, |
| | additional collection of this parameter was |
| | removed as it is not considered necessary for |
| | monitoring of potential liver injury. |
| Cartina to hard | 551255215521 1722 |
| Section to be changed | 5.5.1.2, 5.5.2.1, 5.5.3.1 and 7.3.2 |

c17703547-05 Trial Protocol 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Number of global amendment | 1.0 |
|---|---|
| <b>3</b> | |
| Description of change | Update to include name of metabolite. |
| Rationale for change | The name of metabolite to be measured was |
| _ | added based on the recent data. |
| Section to be changed | 5.2.4.1 |
| Description of change | Clarification on timing and evaluation of triple ECGs. |
| Rationale for change | Clarification |
| Section to be changed | 9.2 References |
| Description of change | Updated reference c02094779-02 to |
| | c02094779-03. |
| | Added missing references R05-0788 and R09- |
| | 4830. |
| Rationale for change | Reference (Investigator brochure) has been |
| | updated since final protocol. |
| Section to be changed | -2.2 |
| | -2.3.2 |
| | -2.3.3 |
| | -4.1.3 |
| | -5.2.5.1 |
| | -5.5.3.1 |
| | -6.2.2 |
| D : 4: 6.1 | -Appendix 10.1 |
| Description of change | -BI1015550 typo corrected |
| | -typo- know corrected to known |
| | - 'one' corrected to 'on' and duplicate word 'patient' removed |
| | -typo in half-life corrected (16-29 hours) was |
| | incorrectly listed as (2016 -29) |
| | -reference to ear removed as oral temperature is |
| | required |
| | 1 dansa |
| | -removed duplicate wording 'or relocate to a |
| | nearby facility overnight' |
| | -deleted typo 'o' |
| Rationale for change | Correction of typos |
| | / 1 |

c17703547-05

**Trial Protocol** 


| Number of global amendment | 2.0 |
|---|---|
| Date of CTP revision | 06 Dec 2018 |
| EudraCT number | 2017-002736-16 |
| BI Trial number | 1305-0012 |
| BI Investigational Product(s) | BI 1015550 |
| Title of protocol | Safety, tolerability, and pharmacokinetics of multiple rising oral doses of BI 1015550 in |
| | patients with idiopathic pulmonary fibrosis (IPF) on no background anti-fibrotic (Part 1) and safety and tolerability of BI 1015550 on top of |
| | Nintedanib and Pirfenidone (Part 2) |
| | (1 wit 2) |
| To be implemented only after | |
| approval of the IRB / IEC / | |
| Competent Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | |
| IRB / IEC / Competent | |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | |
| 1 1 | |
| Section to be changed | Synopsis |
| Description of change | Main criteria for inclusion. Part 1 SOC |
| | requirements updated for consistency with |
| | changes to exclusion 20 made in global |
| | amendment 1. |
| Rationale for change | Correction |
| 0 | • |
| Section to be changed | Flow chart 1A and 2A |
| Description of change | Weight measurement updated for consistency |
| 1 | between part1 and part 2. Baseline weight |
| | measurement added. |
| Rationale for change | Correction. |
| | • |
| Section to be changed | Flow chart 1A |
| Description of change | <u> </u> |


| Number of global amendment | 2.0 |
|---|---|
| , and the second | evening dose. |
| Rationale for change | Clarification of meaning of "post dose" sample at part 1 EOT visit. As there is no dose taken on day 84 the last dose is taken the evening of day 83. |
| Section to be changed | Flow chart 2A |
| Description of change | Footnote 16 updated to clarify, at day 28 sample to be taken ~12h post day 27 evening dose. |
| Rationale for change | Clarification of meaning of "post dose" sample at part 2 EOT visit. As there is no dose taken on day 28, the last dose is taken the evening of day 27. |
| Section to be changed | 3.3 Exclusion Criteria |
| Description of change | Exclusion 22 "positive testing for fecal calprotectin" has been removed. |
| Rationale for change | Calprotectin is a stable protein released by white blood cells during inflammation. Fecal Calprotectin (FC) constitutes an unspecific biomarker of gastrointestinal inflammation. A considerable variability among measurements in the same fecal sample or different samples from stools of consecutive days of the same patient is possible [R16-1924]. FC is established in general practice to only help clinicians differentiate between Irritable Bowel Syndrome (IBS) and Inflammatory Bowel Disease (IBD) in the presence of suspicious symptoms, or in the ongoing monitoring of established IBD. It is not established for any other purpose. Experience in the first IPF cohort of this study shows unexpectedly high baseline values (average above 50 mcg/g) together with a very high intrapatient variability also without drug treatment (with changes of up to 10 fold), independent of any GI symptoms or changes in other laboratory parameters. FC is increased with increase age, concomitant diseases such as GERD, colonic polyps, diabetes, and concomitant medications such as NSAIDs and PPIs. The high frequency of such |

**Trial Protocol** 

| Name to a Calabata | 2.0 |
|---|---|
| Number of global amendment | 2.0 |
| | concomitant diseases and medications in IPF and in the elderly population highly contribute to FC fluctuations. As FC has not been systematically evaluated in IPF, an influence of the underlying disease cannot be excluded. |
| | Overall, given the high variability in the measure in this population within and between patients, also independent of study medication and multiple underlying reasons for increase, the utility of FC cut off values for inclusion in the current study is not appropriate. |
| | Consequently, FC will no longer be considered an exclusion criterion in this trial. FC will continue to be measured at the specified time points in the trial, to allow an exploratory analysis. |
| | Investigator judgment on the overall clinical picture will continue to apply during the study. |
| Section to be changed | 5.2.5.3 |
| Description of change | Information added to standardize weight measurements |
| Rationale for change | To ensure consistency and minimize variability in weight due to time of day or clothing. |
| Section to be changed | 9.2 References |
| Description of change | Gisbert 2009 reference added [R16-1924] |
| Rationale for change | New reference. |
| | New reference. |

c17703547-05 **Trial Protocol** 

| Number of global amendment | 3.0 |
|---|---|
| Date of CTP revision | 12 Feb 2019 |
| EudraCT number | 2017-002736-16 |
| BI Trial number | 1305-0012 |
| BI Investigational Product(s) | BI 1015550 |
| Title of protocol | Safety, tolerability, and pharmacokinetics of multiple rising oral doses of BI 1015550 in patients with idiopathic pulmonary fibrosis (IPF) on no background anti-fibrotic therapy. |
| To be implemented only after approval of the IRB / IEC / Competent Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | |
| IRB / IEC / Competent | |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | |
| Section to be changed | Cover page, Synopsis |
| Description of change | Title, lay title |
| Rationale for change | Updated to reflect removal of part 2 (on top of standard of care) |
| | standard of care) |
| Section to be changed | Cover page, Section 3.1.1, 3.3.5, |
| Description of change | Trial clinical monitor updated to Clinical trial |
| Description of change | leader |
| Rationale for change | For consistency with updated Boehringer |
| in the same of the | Ingelheim trial team titles. |
| 1 | |
| Section to be changed | Synopsis, Flow chart (2a, b, c), Section 2, Section |
| | 3 (including figure 3.1:1 and 3.1:2), Section 4, |
| | Section 5, Section 6, Section 7 |
| Description of change | All references to part 2 – BI 1015550 on top of |
| | SOC have been removed. Terminology stating |
| | Part 1 has removed as no longer required. |
| Rationale for change | Part 2 'BI 1015550 on top of standard of care' is |
| | no longer planned to be conducted within this |
| | phase 1C trial. A short treatment duration of 4 |

**Trial Protocol** 


| Number of global amendment | 3.0 |
|---|---|
| <b>S</b> • | weeks is not adequate to support efficacy or |
| | biomarker endpoints given recent data from the |
| | INMARK trial (1199.227), and therefore removal |
| | of part 2 helps to focus the study from a logistic |
| | and practical point of view on safety and |
| | tolerability and pharmacodynamics of BI |
| | 1015550 in a treatment naïve population. |
| • | |
| Section to be changed | Synopsis, Section 3.3, section 7.6 |
| Description of change | Number of patients has been updated from 36 to |
| | 18 |
| Rationale for change | Result of removal of part 2, only 18 treatment |
| | naïve patients will be recruited. |
| | • |
| Section to be changed | Section 1.2.4, 2.3.2, 3.1.1, 4.1.4.3, 4.2.1, section |
| | 5, section 6.2.2 |
| Description of change | References to nintedanib and pirfenidone or |
| | standard of care (SOC) (within the context of the |
| | removal of study part 2) have been removed. |
| Rationale for change | See rationale for removal of part 2, above. |
| | • |
| Section to be changed | Synopsis: Duration of treatment |
| <b>Description of change</b> | Changed from 12 weeks to 4 weeks for treatment |
| | naïve patients. |
| Rationale for change | Consistency with change in treatment period. |
| | See rationale for change section 3.2 Discussion of |
| | trial design, including choice of control group |
| Section to be changed | Synopsis: Criteria for safety |
| Description of change | Primary endpoint changed from 12 weeks to on |
| | treatment AEs, for treatment naïve patients. |
| Rationale for change | To allow primary endpoint analysis for all |
| | patients whether at 4 weeks for new patients or 12 |
| | weeks for completed (treatment naïve) patients. |
| Section to be changed | Synopsis: Criteria for safety |
| Description of change | <del> </del> |
| Rationale for change | |
| | <del>_</del> |
| | [F1 |
| Section to be changed | Flow chart 1A: overview |
| Description of change | Visits 10, 11, 12 removed |
| | Visit 9 updated to include EOT (end of treatment) |

**Trial Protocol** 


| Number of global amendment | 3.0 |
|---|---|
| | procedures |
| | "Visit 13/End of Trial" renamed to "End of Trial" |
| Rationale for change | With change in treatment duration, visits after day |
| | 28 visit 9 are no longer required. |
| Section to be changed | Flow chart 1A: Footnote 13 and 15 |
| Description of change | Requirements updated in consideration of new |
| | treatment duration. |
| Rationale for change | Requirement for sampling for PK |
| | updated to remove samples past day 28. |
| Section to be changed | 1.2.5.1 Clinical Safety |
| Description of change | Information on completed and ongoing trials has |
| | been updated. New references have been added. |
| Rationale for change | Trial results have become available since initial |
| _ | protocol and have been updated accordingly. |
| | Information on additional trials in program (1305- |
| | 0015 and 1305-0017) have been added. |
| _ | |
| Section to be changed | 1.2.5.1.3 SRD and MRD Study |
| Description of change | Addition of weight data from study 1305.11 |
| Rationale for change | For completion with final study report of 1305.11 |
| Section to be changed | Tables 1.2.5.2.1:1 and 1.2.5.2.2:1 |
| Description of change | Updated results |
| Rationale for change | Consistent with final study report for 1305.11 |
| Section to be changed | 1.2.5.2.1 Single rising dose trial |
| Description of change | Statement 'data from 1305-0011 are preliminary' |
| | has been removed |
| | Data updated based on final report. |
| Rationale for change | Data are no longer preliminary as trial is |
| | complete. Updated values based on final report. |
| | 1050004141 |
| Section to be changed | 1.2.5.2.2 Multiple rising dose trial |
| Description of change | Final report pending removed and reference |
| D 4: 1 C 1 | added. |
| Rationale for change | Final report is now available |
| Cartan ta ba aba | 1 2 5 2 2 Ear 1 offered toil-1 |
| Section to be changed | 1.2.5.2.3 Food effect trial |
| Description of change | Reference added. |
| Rationale for change | Based on final report. |
| | 220 64 1 |
| Section to be changed | 2.3 Benefit risk assessment |


| Number of global amendment | 3.0 |
|---|---|
| Description of change | Rewording regarding target engagement in |
| Description of change | completed study 1305.11 |
| Rationale for change | Consistency with final report |
| Trationale for enange | Consistency with final report |
| Section to be changed | 2.3 Benefit risk assessment |
| Description of change | References to 1305-0011 are updated from |
| Description of change | preliminary and statement regarding TE |
| | biomarkers added. |
| Rationale for change | Information now based on final report. |
| Rationale for change | information now based on final report. |
| Cooking to be about d | 2.3 Benefit risk assessment |
| Section to be changed | _ |
| Description of change | Update of treatment period from 12 to 4 weeks. |
| Rationale for change | Consistency with change in treatment period. |
| | See rationale for change section3.2 Discussion of |
| | trial design, including choice of control group |
| Section to be changed | 3.1 Overall trial design and plan & |
| | Figure 3.1:1 1305-0012 study design overview |
| | Figure 3.1:2 Design and decision point |
| Description of change | Updated references to treatment period from 12 to |
| | 4 weeks. |
| Rationale for change | Consistency with change in treatment period. |
| | See rationale for change section 3.2 Discussion of |
| | trial design, including choice of control group |
| Section to be changed | 3.1.1 Administrative structure |
| Description of change | Updated number of trial sites to approximately 20 |
| Rationale for change | Trial site participation has been expanded to |
| | include additional sites as needed to support |
| | recruitment. |
| | 228: |
| Section to be changed | 3.2 Discussion of trial design, including choice of |
| | control group |
| Description of change | Rationale included supporting reduction of |
| | treatment duration from twelve to four weeks. |
| Rationale for change | Non clinical toxicology data currently supports |
| | studies up to 12 weeks of durations. A treatment |
| | duration of 4 weeks however, is sufficient to |
| | capture safety and tolerability of a PDE4 inhibitor |
| | in support of longer term studies, evaluate PK and |
| | explore induction potential, |
| | in a patient population. |
| | Disease specific biomarkers and pulmonary |
| | function outcomes would require longer than 4 |
| | ranction outcomes would require longer than 4 |


| Number of global amendment | 3.0 |
|---|---|
| | weeks. Recent disease specific biomarker data from the INMARK study (1199-0227) suggest that effects on disease specific exploratory biomarkers would require much larger sample size and with longer duration, to gain a robust evaluation of disease specific biomarkers. Four weeks data allows first generation of normative data on BI 1015550. |
| Section to be changed | 3.3.2 Inclusion criteria |
| Description of change | Inclusion 6 removed |
| Rationale for change | No longer relevant with removal of study part 2 (SOC) |
| Section to be changed | 4.1.1 Identity of BI investigational product and comparator product |
| Description of change | Duration of use updated from 84 days to 28 days for both BI 1015550 and Placebo matching. |
| Rationale for change | Consistency with change in treatment period. See rationale for change section 3.2 Discussion of trial design, including choice of control group |
| Section to be changed | 4.1.3 Selection of doses in the trial |
| Description of change | Information regarding 1305-0011 trial was updated to final. Rewording of starting dose justification. |
| Rationale for change | Information now based on final report. |
| Section to be changed | 4.1.4.2 Dispensing of medication |
| Description of change | Table 4.1.4.2:1 Quantity of medication kits dispensed per visit |
| Rationale for change | Updated based on revised treatment duration and visit schedule. |
| Section to be changed | 4.1.4.3 Administration of dose |
| Description of change | Added "taken at home since last clinic visit" |
| Rationale for change | For clarification on when the diary should be filled in |
| Section to be changed | 5.1.1 Endpoints of Efficacy |
| Description of change | 12 week time point removed from all endpoints as per revised treatment duration. Rewording to "over time" rather than 4 and 12 weeks |
| Rationale for change | To allow PE analysis for all patients whether at 4 |


| Number of global amendment | 3.0 |
|---|---|
| | weeks for new patients or 12 weeks for completed |
| | patients |
| Section to be changed | 5.2.1 Endpoints of safety |
| Description of change | Primary endpoint (for treatment naïve patients) changed to "AEs on treatment" rather than 4 weeks or 12 weeks. To allow PE analysis for all patients whether at 4 weeks for new patients or 12 weeks for completed patients. |
| Rationale for change | Consistency with change in treatment period. See rationale for change section 3.2 Discussion of trial design, including choice of control group |
| Section to be changed | |
| Description of change | † |
| 2 compton of change | |
| Rationale for change | |
| Section to be changed | 6.2.1 Saraaning and run in pariod(s) |
| Section to be changed Description of change | 6.2.1 Screening and run in period(s) Addition of "Screening period may be extended |
| Description of change | for administrative reasons. Approval should be obtained from the sponsor who will also determine if any tests specified in the protocol must be repeated before the randomization visit." |
| Rationale for change | To allow flexibility between screening and pre- |
| | randomisation visit especially when escalating to |
| | the next dose level, hence potential time gap for |
| | safety review of previous cohort |
| Section to be changed | 6.2.2 Treatment period |
| Description of change | Addition of "will be given a diary to record intake |
| | of study medication taken at home since the last |
| Dationals for shangs | visit" To clarify the timing of the recording of the study |
| Rationale for change | To clarify the timing of the recording of the study medication intake since the last visit. |
| | medication make since the last visit. |
| Section to be changed | 6.2.2 Treatment period |
| beenon to be changed | |
| Description of change | * |
| Description of change | End of treatment visit: End of treatment visit timing changed from visit |


| Number of global amendment | 3.0 |
|---|---|
| | patients. Explanation of requirements for EOT visit for prematurely discontinued patients if patients discontinue, changed from 'prior to 12 weeks' to 'prior to 4 weeks'. |
| Rationale for change | Consistency with change in treatment period. See rationale for change section3.2 Discussion of trial design, including choice of control group |
| Section to be changed | 9.0 References |
| Description of change | New references added |
| Rationale for change | New reference. |

c17703547-05 **Trial Protocol**  Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Number of global amendment | 4.0 |
|---|---|
| Date of CTP revision | 27 MAR 2019 |
| EudraCT number | 2017-002736-16 |
| BI Trial number | 1305-0012 |
| BI Investigational Product(s) | BI 1015550 |
| Title of protocol | Safety, tolerability, and pharmacokinetics of multiple rising oral doses of BI 1015550 in patients with idiopathic pulmonary fibrosis (IPF) on no background anti-fibrotic therapy. |
| To be implemented only after approval of the IRB / IEC / Competent Authorities | |
| To be implemented immediately in order to eliminate hazard – IRB / IEC / Competent Authority to be notified of change with request for approval | |
| Can be implemented without IRB / IEC / Competent Authority approval as changes involve logistical or administrative aspects only | |
| Section to be changed | Synopsis Section 3.1 Table 3.1:1 Section 3.2 Section 7.6 |
| Description of change | Information regarding the addition of 6 patients (4 active, 2 placebo) to the 18mg bid dose group, has been added. |
| Rationale for change | Further to the safety review, for the purpose of escalation, of the completed 2 weeks treatment of the 9 patients in the 18 mg bid cohort, whilst safety and tolerability were considered acceptable, the prediction for the 24 mg bid cohort regarding the AUC gMean (2290 nM*h) exceeded the threshold (2284 nM*h) as set in the protocol on the basis of the 13 weeks rat toxicology data. The observed PK data of the 18 mg bid cohort showed a higher variability, including outliers, in IPF patients as compared to the HV data. It is therefore deemed appropriate to |

c17703547-05 **Trial Protocol**  Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| extend the current 18 mg bid cohort (4 on verum and 2 on placebo) to further characterize, understand and refine PK variability at 2 weeks in the target IPF population. Increasing the number of patients may confirm the magnitude of the PK variability. After 6 additional patients, the safety review committee will review all 18mg bid patient data, in order to determine if escalation can proceed to the 24 mg bid cohort. This will only occur if the safety and tolerability are maintained as |
|---|
| acceptable and if PK projections for the next dose are within defined limits. |
| Section 7.3.4 |
| Third paragraph, change in wording "In contrast to final PK calculations, the preliminary analysis will be based on planned sampling times rather than actual times" was changed to "In contrast to final PK calculations, the preliminary analysis may be based on planned sampling times rather than actual times" |
| This modification is made to allow a decision to proceed with analysis using planned times or directly with actual times. As there may be a relevant discrepancy in actual sampling times and planned sampling times, actual times can be preferable in the PK analysis. |



#### APPROVAL / SIGNATURE PAGE

Document Number: c17703547 Technical Version Number: 5.0

**Document Name:** clinical-trial-protocol-version-05

**Title:** Safety, tolerability, and pharmacokinetics of multiple rising oral doses of BI 1015550 in patients with idiopathic pulmonary fibrosis (IPF) on no background anti-fibrotic therapy.

## **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Author-Clinical Trial Leader | | 27 Mar 2019 15:55 CET |
| Author-Trial Statistician | | 27 Mar 2019 15:58 CET |
| Author-Trial Clinical<br>Pharmacokineticist | | 27 Mar 2019 16:02 CET |
| Approval-Team Member Medicine | | 27 Mar 2019 16:31 CET |
| Approval-Therapeutic Area | | 28 Mar 2019 10:16 CET |
| Verification-Paper Signature<br>Completion | | 28 Mar 2019 14:11 CET |

**Boehringer Ingelheim Document Number:** c17703547 **Technical Version Number:**5.0

# (Continued) Signatures (obtained electronically)

| Meaning of Signature Signed by Date Signed |
|--------------------------------------------|
|--------------------------------------------|